Official Title: Study of Nasal Insulin to Fight Forgetfulness - Combination Intranasal Insulin and Empagliflozin Trial

NCT05081219

IRB Approval Date: 07/14/23

## Study of Nasal Insulin to Fight Forgetfulness (SNIFF)

## **SNIFF Combination Intranasal Insulin and Empagliflozin Trial**

## PROJECT DIRECTOR / IND SPONSOR

Suzanne Craft, Ph.D.

Wake Forest University Health Sciences/ Wake Forest School of Medicine
Medical Center Boulevard
Winston-Salem, NC 27157-1207

suzcraft@wakehealth.edu Tel: 336-713-8832

## PROTOCOL VERSION

Final Protocol v5.0 July 14, 2023

# **TABLE OF CONTENTS**

| 1.0 I | NTRODUCTION | 9 |
|---|---|---|
| 1.1 | Primary Aim | |
| 1.2 | Secondary Aim 1 | 10 |
| | CKGROUND AND SIGNIFICANCE | |
| 2.1 | Rationale for Insulin | |
| 2.2 | Insulin as a Therapeutic Agent | |
| 2.3 | Intranasal Pathways to the CNS | 11 |
| 2.4 | Intranasal Delivery System Devices | 12 |
| | ELIMINARY STUDIES | |
| 3.1 | Participants | |
| 3.2 | Procedures | |
| 3.3 | Safety and Compliance | |
| 3.4 | Statistical Analyses | |
| 3.5<br>3.6 | Results: Cognitive and Functional Outcome Measures | |
| 3.6<br>3.7 | Results: AD Biomarkers | |
| 3.8 | | |
| 3.9 | Safety and Compliance | 17 |
| | · | |
| 4.0 <b>PF</b> | ELIMINARY STUDY 2 | 17 |
| 5.0 <b>PF</b> | ELIMINARY STUDY 3 | 19 |
| 5.1 | Rationale for Dosage Selection | 20 |
| 5.2 | Rationale for Primary and Secondary Outcome Measures | 20 |
| 5.3 | Rationale for Design of Trial | |
| 5.4 | Rationale for Biofluids | 20 |
| 6.0 <b>ST</b> | UDY OVERVIEW | 20 |
| 6.1 | Study Population | 20 |
| 6.2 | Diagnosis Criteria | 20 |
| 6.3 | Inclusion Criteria | |
| 6.4 | Exclusion Criteria | |
| 6.5 | Recruitment and Retention Strategies | 22 |
| 7.0 <b>ST</b> | UDY TIMELINE | 22 |
| 8.0 <b>DE</b> | SCRIPTION OF STUDY VISITS | 22 |
| 8.1 | Screening (Visit 1) | |
| 8.2 | Baseline Visit 1 (Visit 2) | |
| 8.3 | Baseline Visit 2 (Visit 3; one week after Baseline Visit 1) | |
| 8.4 | Re-supply Visit and Safety/Compliance Assessment 1 (Visit 4; one week after | |
| 2) | 23 | |
| 8.5 | Phone Safety/Compliance Assessment 2 | 23 |
| 8.6 | Post-treatment Visit 1 (Visit 5) | |
| 8.7 | Post-treatment Visit 2 (Visit 6; one week after Post-treatment Visit 1) | 24 |
| 9.0 <b>ST</b> | UDY-SPECIFIC PROCEDURES | 24 |
| 9.1 | Cognitive Evaluation Instruments Administered to the Participant | |
| 9.2 | Clinical and Functional Evaluations | 24 |
| 9.2.1 | Quick Dementia Rating System (QDRS) | 24 |
| 9.2.2 | Activities of Daily Living Scale for MCI/ADL-MCI | 24 |
| 10 0 <b>ST</b> | UDY METHODS | 25 |

| 10.1 | Safety Assessments | 25 |
|---|---|---|
| 10.2 | Physical and Neurological Examination | |
| 10.3 | Electrocardiogram (ECG) | |
| 10.4 | Clinical Laboratory Evaluations | |
| 10.5 | Actigraphy | |
| 10.6 | Continuous Glucose Monitoring | 25 |
| | DMARKER STUDIES | |
| 11.1 | CSF | |
| 11.2 | Blood Collection at Lumbar Puncture Visits | |
| 11.3 | Genetic Samples, Storage and Future Use | 26 |
| 12.0 <b>ST</b> | ATISTICAL PLAN | 26 |
| 12.1 | Power Analyses | 26 |
| 13 0 <b>PC</b> | TENTIAL RISKS | 26 |
| 13.1 | Safety of Intranasal Insulin | |
| 13.2 | Risks associated with use of the Aptar CPS device | |
| 13.3 | Risks associate with use of the Empatica E4 actigraphy device | |
| 13.4 | Risks associated with use of the Libre Freestyle Pro Glucose Monitoring System | |
| 13.5 | Lumbar Puncture | 28 |
| 13.6 | Blood Draw | 28 |
| 14 0 <b>PF</b> | RSONNEL REQUIREMENTS | 28 |
| | UDY DRUGS | |
| 15.1<br>15.2 | Humulin® R U-100 InsulinRandomization | |
| 15.2 | Blinding | |
| 15.4 | Study Drug Dispensing | |
| 15.5 | Intranasal Administration | |
| 15.6 | Storage | |
| 15.7 | Drug Accountability | |
| 16 O AF | VERSE EVENTS | 30 |
| 16.1 | Definition | |
| 16.2 | Following Up on AEs | |
| 17.0 <b>SE</b><br>17.1 | RIOUS ADVERSE EVENTS (SAE) | |
| 17.1<br>17.2 | Definition Reporting SAEs | |
| 17.2 | IND Safety Reporting | |
| | • • • | |
| | HICS & REGULATORY CONSIDERATIONS | |
| 18.1 | Ethical StandardInstitutional Review Board (IRB) | 31 |
| 18.2<br>18.3 | Informed Consent & HIPAA Authorization | |
| 18.4 | Participant Confidentiality HIPAA | |
| | • | |
| | NETIC RESEARCH & STORAGE OF GENETIC MATERIAL | |
| 19.1 | Storage of Biospecimen Samples | |
| 20.0 <b>RIS</b> | SKS AND BENEFITS ASSOCIATED WITH THIS STUDY | 33 |
| 20.1 | Potential Benefits of the Proposed Research to Human Subjects | 33 |
| 20.2 | Inclusion of Women and Minorities | |
| 20.3 | Inclusion of Children as Participants in Research Involving Human Subjects | |
| 20.4 | Data and Safety Monitoring Plan | 33 |

| 21.0 | PUBLICATION POLICY | 34 |
|------|-------------------------------------------------|----|
| 22.0 | SHARING OF FINAL RESEARCH DATA | 34 |
| 23.0 | TABLE 4: SCHEDULE OF PROCEDURES AND ASSESSMENTS | 35 |
| 24.0 | LITERATURE CITED | 37 |

# STUDY GLOSSARY

| 3MSE | MODIFIED MINI-MENTAL STATUS EXAM |
|---|---|
| AB | BETA AMYLOID |
| AD | ALZHEIMER'S DISEASE |
| ADAS-COG | ALZHEIMER'S DISEASE ASSESSMENT SCALE – COGNITIVE SUBSCALE |
| ADCS | ALZHEIMER'S DISEASE COOPERATIVE STUDY |
| ADCS-ADL | ALZHEIMER'S DISEASE COOPERATIVE STUDY - ACTIVITIES OF DAILY LIVING |
| ADEAR | ALZHEIMER'S DISEASE EDUCATION AND REFERRAL CENTER |
| ADNI | ALZHEIMER'S DISEASE NEUROIMAGING INITIATIVE |
| AE | ADVERSE EVENT |
| AMCI | AMNESTIC MILD COGNITIVE IMPAIRMENT |
| ANCOVA | ANALYSIS OF COVARIANCE |
| APOE/APOE4 | APOLIPOPROTEIN (APOE) EPSILON 4 (APOE4) |
| BDNF | BRAIN-DERIVED NEUROTROPHIC FACTOR |
| BID BID | BIS IN DIE (TWICE A DAY) |
| BUN | BLOOD UREA NITROGEN |
| CDR-SB | CLINICAL DEMENTIA RATING – SUM OF BOXES |
| CFR | CODE OF FEDERAL REGULATIONS |
| CMRGLC | CEREBRAL METABOLIC RATE OF GLUCOSE UTILIZATION |
| CNS | CENTRAL NERVOUS SYSTEM |
| CPD | CONTROLLED PARTICLE DISPERSION |
| СРК | CREATINE PHOSPHOKINASE |
| CREB | CAMP RESPONSE ELEMENT-BINDING PROTEIN |
| CRF/E-CRF | CASE REPORT FORM/ELECTRONIC CASE REPORT FORM |
| CSF | CEREBRAL SPINAL FLUID |
| DNA | DEOXYRIBONUCLEIC ACID |
| DSMB | DATA & SAFETY MONITORING BOARD |
| DSM-IV | DIAGNOSTIC AND STATISTICAL MANUAL OF MENTAL DISORDERS, FOURTH EDITION |
| DSRS | DEMENTIA SEVERITY RATING SCALE |
| EAG | ESTIMATED AVERAGE GLUCOSE |
| ECG | ELECTROCARDIOGRAM |
| EDC | ELECTRONIC DATA CAPTURE |

| EDTA | ETHYLENE DIAMINE TETRA ACETIC ACID |
|---------|-----------------------------------------------------|
| ELISA | ENZYME-LINKED IMMUNOSORBENT ASSAY |
| EMPA | EMPAGLIFLOZIN |
| FCSRT | FREE AND CUED SELECTIVE REMINDING TEST |
| FDA | FOOD AND DRUG ADMINISTRATION |
| FDG PET | FLUORO DEOXY GLUCOSE POSITRON EMISSION TOMOGRAPHY |
| GCP | GOOD CLINICAL PRACTICE |
| GEE | GENERALIZED ESTIMATING EQUATION |
| GGT | GAMMA GLUTAMYL TRANSPEPTIDASE |
| GSK3B | GLYCOGEN SYNTHASE KINASE 3 BETA |
| HGA1C | HEMOGLOBIN A1C |
| НС | HOMOCYSTEINE |
| нст | HEMATOCRIT |
| НСҮ | HOMOCYSTEINE |
| HEENT | HEAD EARS EYES NOSE THROAT |
| HGB | HEMOGLOBIN |
| HIPAA | HEALTH INSURANCE PORTABILITY AND ACCOUNTABILITY ACT |
| HOMA-IR | HOMEOSTATIS MODEL ASSESSMENT OF INSULIN RESISTANCE |
| ICF | INFORMED CONSENT FORM |
| ICH | INTERNATIONAL CONFERENCE ON HARMONISATION |
| IDE | INSULIN DEGRADING ENZYME |
| IGF-1 | INSULIN-LIKE GROWTH FACTOR-1 |
| INI | INTRANASAL INSULIN |
| IRB | INSTITUTIONAL REVIEW BOARD |
| ITT | INTENT-TO-TREAT |
| LDH | LACTATE DEHYDROGENASE |
| LP | LUMBAR PUNCTURE |
| LTP | LONG TERM POTENTIATION |
| MCV | MEAN CORPUSCULAR VOLUME |
| ML | MILLILITER |
| MMA | METHYLMALONIC ACID |
| MMSE | MINI MENTAL STATE EXAMINATION |
| MPRAGE | MAGNETIZATION PREPARED RAPID GRADIENT ECHO |
| MR/MRI | MAGNETIC RESONANCE / MAGNETIC RESONANCE IMAGING |

| NBAC | NATIONAL BIOETHICS ADVISORY COMMISSION |
|---|---|
| NIA | NATIONAL INSTITUTE ON AGING |
| NIH | NATIONAL INSTITUTES OF HEALTH |
| NINCDS/ADRDA | NATIONAL INSTITUTE OF NEUROLOGICAL AND COMMUNICATIVE DISEASES AND STROKE / ALZHEIMER'S DISEASE AND RELATED DISORDERS ASSOCIATION |
| NBDA | N-METHYL - D-ASPARTATE |
| NSAID | NON-STEROIDAL ANTI-INFLAMMATORY DRUGS |
| OHRP | OFFICE FOR HUMAN RESEARCH PROTECTIONS |
| РВМС | PERIPHERAL BLOOD MONONUCLEAR CELL |
| PD | PROJECT DIRECTOR |
| PCP | PRIMARY CARE PHYSICIAN |
| PET | POSITRON EMISSION TOMOGRAPHY |
| PHI | PROTECTED HEALTH INFORMATION |
| PI | PRINCIPAL INVESTIGATOR |
| PID | PARTICIPANT ID |
| RBC | RED BLOOD CELL |
| RE | RANDOM EFFECTS |
| ROI | REGIONS OF INTEREST |
| SAE | SEVERE ADVERSE EVENT |
| SD | STANDARD DEVIATION |
| SGOT | SERUM GLUTAMIC OXALOACETIC TRANSAMINASE |
| SGPT | SERUM GLUTAMIC PYRUVIC TRANSAMINASE |
| Т | TESLA |
| TSH | THYROID STIMULATING HORMONE |
| U/A | URINALYSIS |
| WBC | WHITE BLOOD COUNT |

| TITLE | Study of Nasal Insulin to Fight Forgetfulness "SNIFF" –<br>Combination Intranasal Insulin and Empagliflozin Trial |
|---|---|
| PROJECT DIRECTOR | Suzanne Craft, Ph.D. |
| STUDY SPONSOR | Wake Forest University Health Sciences (WFUHS) /<br>Alzheimer's Disease Research Center (ADRC) |
| STUDY PHASE | Phase II Pilot Study |
| INDICATION | Preclinical AD, amnestic mild cognitive impairment (aMCI) or mild Alzheimer's disease (AD) |
| AIM OF STUDY | The proposed pilot study will provide safety and efficacy preliminary data regarding singular and combined effects of two therapeutic approaches, intranasal insulin and treatment with the sodium-glucose cotransporter type 2 inhibitor (SGLT2i) empagliflozin, to correct bioenergetic and vascular dysfunction in adults with preclinical AD and amnestic mild cognitive impairment (aMCI) or early AD |
| PRIMARY OBJECTIVE | We will test the hypothesis that 1 month of treatment with INI (40 IU q.i.d.), with the SGLT2i empagliflozin (empa; 10 mg q.d.), and with combined insulin plus empagliflozin (INI+empa) will result in safety profiles (number of treatment-related serious adverse events/primary outcome) that are similar to placebo. |
| SECONDARY OBJECTIVES | We will determine the effects of singular and combined therapy<br>on AD cerebrospinal fluid biomarkers, cerebral blood flow<br>(CBF) and cognition. |
| PRIMARY OUTCOME MEASURE | Number of treatment-related serious adverse events |
| SECONDARY OUTCOME MEASURES | PACC5, ADAS-Cog14, CSF Aβ40, Aβ42, total tau, and phospho-tau 181, whole brain CBF |
| STUDY DESIGN | Single-site, double-blind study |
| SAMPLE SIZE | n=60 |
| SUMMARY OF KEY ELIGIBILITY CRITERIA | <ul> <li>Cognitively normal with positive amyloid (amyloid PET SUVR&gt;1.21, CSF Aβ42&lt;600 pg/ml)</li> <li>Diagnosis of amnestic mild cognitive impairment (MCI) or early AD (CDR 0.5 or 1, MMSE&gt;21)</li> <li>Age: 55 to 85 years (inclusive)</li> </ul> |
| DRUG DOSAGE & FORMULATION | 40 International Units Humulin® R U-100 (Eli Lilly, Inc.) q.i.d.; empagliflozin (10 mg q.d.) |
| DURATION OF PARTICIPATION | 8 weeks (4 weeks on active treatment) |
| PLACEBO | Insulin diluent (Eli Lilly, Inc.); cellulose capsule |

| ROUTE OF ADMINISTRATION | Intranasal (insulin); oral (empagliflozin) |
|---|---|
| PROCEDURES | Physical and neurological exam, nasal examination, cognitive testing, magnetic resonance imaging (MRI), continuous glucose monitoring, actigraphic sleep assessment, lumbar puncture, vitals, clinical labs, CSF and blood analysis and banking and APOE genotyping. |

#### 1.0 INTRODUCTION

An urgent need exists to find effective treatments for AD that can arrest or reverse the disease at its earliest stages. The emotional and financial burden of AD to patients, family members, and society is enormous, and is predicted to grow exponentially as the median population age increases. Current FDA-approved therapies are modestly effective at best. The proposed study will examine singular and combined effects of two novel therapeutic approaches to correct bioenergetic and vascular dysfunction in adults with amnestic mild cognitive impairment (aMCI). Metabolic and vascular disorders are well-known risk factors for Alzheimer's disease (AD); although the mechanisms through which they influence risk is not completely understood, accruing research has identified numerous potential contributors, including insulin resistance, bioenergetic defects, inflammation, impaired vascular function, and reduced clearance of protein aggregates, all of which have cumulative adverse effects on brain function with aging. Based on this evidence, it has been suggested that medications used to treat metabolic and vascular function could be repurposed as therapies for AD.

Sodium-glucose co-transporter-2 inhibitors (SGLT2is) belong to a new class of agents that has attracted considerable interest because of concomitant effects on metabolism and vascular function in adults with Type 2 diabetes and/or cardiovascular disease. In the periphery, SGLT2is reduce hyperglycemia through off-loading of glucose into urine, and modulate sodium handling leading to reduced blood pressure and improved cardiovascular function. They have been tested in numerous large trials and shown to be safe; because they do not increase insulin, they can be administered without risk of hypoglycemia in non-diabetic adults. SGLT2 has been identified in brain, as well as in choroid plexus epithelial cells where it may play a role in cerebrospinal fluid (CSF) production and brain glymphatics. SGLT2 expression in brain is increased with traumatic brain injury and cerebral ischemia. Preclinical studies indicate effects of SGLTis in the brain that are of relevance to AD, including a shift from glycolysis to fatty acid metabolism, thereby providing an alternative energy substrate, enhanced mitochondrial function, decreased oxidative stress, and inhibition of the mTOR signaling pathway. In an AD mouse model, the SGLT2 inhibitor empagliflozin reduced amyloid plagues, inflammation, and microhemorrhages, while enhancing performance on memory measures.

Another approach to correcting brain metabolic and vascular dysregulation in AD involves direct provision of insulin to the brain via intranasal insulin (INI) administration using devices specialized for nose-to-brain delivery. In pilot and Phase II trials this approach improved cerebral glucose utilization, AD CSF biomarker profiles, white matter hyperintensity volume progression, and cognition. Although a recent Phase II trial showed improvement with only one of two devices, in subsequent pilot studies we have determined that this failure may have been due in part to different methods of delivery used by the two devices, requiring different dosing strategies, and have validated a dosing protocol that verifies reliable delivery of insulin to the CNS.

SGLT2is and insulin exert beneficial metabolic and vascular effects in brain through different mechanisms. SGLT2i effects are not directly related to insulin, although through promoting a switch to fatty acid metabolism, peripheral hyperinsulinemia is reduced with corresponding decrease in insulin resistance. In contrast, insulin likely works directly through its receptors which are prolific throughout brain to promote synaptic viability, neurogenesis, and vasoreactivity, with downstream amelioration of amyloid and tau pathology. Thus, although each approach could be predicted to benefit AD symptoms and pathology, it is possible that additive or synergistic effects would be observed by combining the

two approaches. In large trials, insulin and SGLT2is have been co-administered with no adverse events. Further, because intranasal insulin does not lower blood glucose, and SGLT2is lower blood glucose only in the presence of hyperglycemia, and are not associated with hypoglycemia, the combined regimen is likely to be safe. This hypothesis will be tested in the proposed proof of concept study which will examine whether the safety profiles of 4 weeks of combined and singular administration of intranasal insulin and empagliflozin compared with placebo. We will also examine effects of treatment on cognition, CSF biomarkers, and cerebral perfusion. If successful, information gained from the study will inform the design of a future Phase II trial.

## 1.1 **Primary Aim**

We will test the hypothesis that 4 months of treatment with INI (40 IU q.i.d.), with the SGLT2i empagliflozin (empa; 10 mg q.d.), and with combined insulin plus empagliflozin (INI+empa) will result in safety profiles (number of treatment-related serious adverse events/primary outcome) that are similar to placebo.

## 1.2 **Secondary Aim 1**

We will determine the effects of singular and combined therapy on AD cerebrospinal fluid biomarkers, cerebral blood flow (CBF) and cognition.

## 2.0 BACKGROUND AND SIGNIFICANCE

#### 2.1 Rationale for Insulin

The rationale for the study is derived from growing evidence that insulin carries out multiple functions in the brain, and that insulin dysregulation may contribute to AD pathogenesis (Craft and Watson 2004). Insulin receptors are densely localized in the hippocampus and in entorhinal, frontal, and other cortical areas; they are found primarily in synapses, where insulin signaling modulates synaptogenesis and synaptic remodeling (Chiu, Chen et al. 2008, Zhao and Townsend 2009). Insulin facilitates memory at optimal levels, possibly through synaptic effects and enhanced hippocampal glucose utilization (Grillo, Piroli et al. 2009).

The importance of insulin in normal brain function is underscored by evidence that insulin dysregulation contributes to the pathophysiology of AD, a disorder characterized in its earliest stages by synaptic loss and memory impairment. Hoyer and colleagues first identified a reduction in insulin receptors and signaling markers in the AD brain (Frolich, Blum-Degen et al. 1998). This initial finding has been confirmed and extended by other investigators, who have demonstrated reduced CSF insulin in patients with AD and MCI (Craft, Peskind et al. 1998, Gil-Bea, Solas et al. 2010), and reduced insulin and IGF-I messaging with increasing AD pathology and cholinergic deficit (Rivera, Goldin et al. 2005). Insulin has a close relationship with β-amyloid, the toxic peptide produced by cleavage of the amyloid precursor protein (Zhao and Townsend 2009). In AD, insoluble Aß peptides deposit in brain parenchyma and vasculature. Soluble Aβ species, particularly oligomers of the 42 amino acid specie (Aβ42), have synaptotoxic effects, possibly resulting in synapse loss, which is the earliest structural defect observed in AD (Selkoe 2008). Insulin reduces oligomer formation and protects against Aβ-induced synaptotoxicty and LTP disruption (Gasparini, Gouras et al. 2001, De Felice, Vieira et al. 2009, Lee, Kuo et al. 2009). Interestingly, Aβ also regulates brain insulin signaling. Soluble A\( \beta \) binds to the insulin receptor and disrupts insulin signaling and LTP induction in mouse hippocampal slice preparations (Townsend, Mehta et al. 2007). These effects could be prevented by exposing tissue to insulin prior to Aβ exposure. Insulin pre-treatment also prevented synthetic soluble Aβ oligomers from downregulating plasma membrane insulin receptors and reducing dendritic spines in primary hippocampal neurons (De Felice, Vieira et al. 2009). Insulin may also modulate Aß degradation by regulating expression of insulin degrading enzyme (IDE), a metalloprotease that catabolizes insulin (Zhao, Teter et al. 2004). Collectively, these findings suggest that soluble Aβ may

induce central nervous system (CNS) insulin resistance and synapse loss, and that treatment with insulin may prevent these pathological processes.

A role for insulin has also been suggested for other AD-related mechanisms. Insulin inhibits phosphorylation of tau, through its regulation of glycogen synthase kinase  $3\beta$ , a downstream target in the insulin signaling pathway (Hong and Lee 1997). Insulin dysregulation is also associated with oxidative stress, inflammation, and impaired neurogenesis (Craft and Watson 2004). Thus, insulin has been implicated in numerous processes related to AD pathophysiology, suggesting that correction of insulin dysregulation may be a therapeutic strategy with considerable clinical and scientific significance.

## 2.2 Insulin as a Therapeutic Agent

The study uses insulin as a therapeutic agent and intranasal administration focusing on nose to brain transport as a mode of delivery. As reviewed above, insulin has pleiotropic effects on pathways implicated in AD pathogenesis. As such, augmenting CNS insulin is an alternative approach to AD therapy, in contrast to the majority of therapeutic approaches that focus on narrowly defined mechanisms such as acetylcholine modulation or amyloid accumulation. Restoring normal brain insulin levels in persons with AD may improve cognition and AD pathologic processes. Such an approach is possible with an intranasal administration technique.

## 2.3 Intranasal Pathways to the CNS

Olfactory sensory neurons are directly exposed to the external environment in the upper nasal cavity while their axons extend through the cribriform plate to the olfactory bulb. Following intranasal administration, drugs can be directly transported to the CNS, bypassing the periphery. Several extraneuronal and intraneuronal pathways from the nasal cavity to the CNS are possible. The extraneuronal pathways appear to rely on bulk flow transport through perineural channels to the brain or CSF. In recent studies, labeled INI or a closely related peptide, insulin-like growth factor-I (IGF-I). were administered to rodents (Thorne, Pronk et al. 2004, Francis, Martinez et al. 2008). Within 30 minutes, signal was detected along olfactory and trigeminal channels, as well as in the hippocampus, amygdala and rostral and caudal cortex. An additional extracellular pathway was identified with guick access to the CSF after absorption into the submucosa along the olfactory nerve and cribriform plate (Born, Lange et al. 2002, Frey 2002, Thorne, Pronk et al. 2004). These extracellular pathways provide direct access to the CNS within minutes of intranasal administration. Additionally, an intraneuronal pathway delivers drugs to the CNS hours or days later (Broadwell and Balin 1985, Shipley 1985, Baker and Spencer 1986, Balin, Broadwell et al. 1986). Viruses and microorganisms (Fairbrother and Hurst 1930, Faber 1938, Bodian and Howe 1941), amino acids (Weiss and Holland 1967), and proteins (Kristensson and Olsson 1971, Shipley 1985, Thorne, Emory et al. 1995) can also enter the CNS via nasal routes. In particular, substances with lower molecular weights are more likely to be transported to the CNS along intranasal pathways (Sakane, Akizuki et al. 1995). Insulin's molecular weight of about 5800 g/mol makes it a good candidate for intranasal delivery. Animal studies show labeled uptake to hippocampus and rostral and caudal cortex following INI administration (Francis, Martinez et al. 2008). In a murine diabetes model, INI reduced brain atrophy, while increasing synaptic markers and activation of Akt, CREB, and GSK3β. Memory enhancement was also observed on Water Maze and radial arm tasks (Francis, Martinez et al. 2008). Human functional and cognitive studies of INI also support insulin's transport to the CNS. INI treatment increases CSF insulin levels and induces changes in auditory-evoked brain potentials compared to placebo (Kern, Born et al. 1999). INI improves verbal memory acutely in persons with AD and aMCI without affecting plasma insulin or glucose levels at the dose included in the study (Reger, Watson et al. 2006). Regarding chronic effects, several studies reported that 2 months of daily insulin administration (160 International Units/day) significantly improves verbal memory in young healthy adults (Benedict, Hallschmid et al. 2004, Stockhorst, de Fries et al. 2004, Benedict, Kern et al. 2008, Hallschmid, Benedict et al. 2008, Stockhorst, de Fries et al. Submitted for publication). Finally, Section 3.0 presents results in a

preliminary study in which insulin was administered to adults with AD or aMCI for 4 months.

## 2.4 Intranasal Delivery System Devices

The intranasal delivery device to be used in this study has been developed and extensively tested by Aptar Pharmaceuticals, a company specializing in drug delivery. Specifications and instructions for the device are provided in attached materials:

1) The CPS pump is a multidose device utilizing an air-filtered preservative free system, in which a .2 micrometer filter membrane filters the airflow and insulin will be delivered through a spring loaded tip. This device is currently used in the delivery of Esketamine, a Janssen product approved by the FDA for the treatment of refractory depression.

# 2.5 Rationale for Sodium-Glucose Cotransporter Type 2 Inhibitors for the Treatment of Alzheimer's Disease

As noted previously, metabolic and vascular disorders are well-known risk factors for Alzheimer's disease (AD); although the mechanisms through which they influence risk is not completely understood, accruing research has identified numerous potential contributors, including insulin resistance, bioenergetic defects, inflammation, impaired vascular function, and reduced clearance of protein aggregates, all of which have cumulative adverse effects on brain function with aging. Based on this evidence, it has been suggested that medications used to treat metabolic and vascular function could be repurposed as therapies for AD.

Sodium-glucose co-transporter-2 inhibitors (SGLT2is) belong to a new class of agents that has attracted considerable interest because of concomitant effects on metabolism and vascular function in adults with Type 2 diabetes and/or cardiovascular disease. In the periphery, SGLT2is reduce hyperglycemia through off-loading of glucose into urine, and modulate sodium handling leading to reduced blood pressure and improved cardiovascular function. They have been tested in numerous large trials and shown to be safe; because they do not increase insulin or lower glucose except in the context of hyperglycemia, they can be administered without risk of hypoglycemia in non-diabetic adults. SGLT2 has been identified in brain, as well as in choroid plexus epithelial cells where it may play a role in cerebrospinal fluid (CSF) production and brain glymphatics. SGLT2 expression in brain is increased with traumatic brain injury and cerebral ischemia. Preclinical studies indicate effects of SGLTis in the brain that are of relevance to AD, including a shift from glycolysis to fatty acid metabolism, thereby providing an alternative energy substrate, enhanced mitochondrial function, decreased oxidative stress, and inhibition of the mTOR signaling pathway. In an AD mouse model, the SGLT2 inhibitor empagliflozin reduced amyloid plaques, inflammation, and microhemorrhages, while enhancing performance on memory measures.

Empagliflozin has been tested in large trials of patients with Type 2 diabetes and cardiovascular disease (i.e., EMPA-REG OUTCOME) and like other SGLT2is has been shown to have an excellent safety profile (as reviewed in Scheen, Nature, 2020), improving glucose metabolism and reducing the incidence of major cardiovascular events. Adverse events that occur infrequently include diabetic ketoacidosis and genital infection. Medical monitoring for the study will be carried out by an experienced diabetologist, Don McClain, MD, and by a neurologist expert in care of adults with Alzheimer's disease, James Trey Bateman, MD, MPH.

#### 3.0 PRELIMINARY STUDIES

A preliminary study examined the impact of 4-month INI administration using the ViaNase device (10 or 20 International Units bid vs. placebo) on the primary outcome measures of delayed story recall and the Dementia Severity Rating Scale (DSRS) as well as on measures of global cognition and function used in traditional AD clinical trials. In a subset of participants, effects on CSF AD biomarkers

(Aβ42 and tau/Aβ42 ratio), and on cerebral metabolic rate of glucose utilization (CMRglc) assessed by F18FDG PET were also examined (Craft, Baker et al. 2012).

## 3.1 Participants

A total of 111 older adults were randomized in the study (Fig. 1). Data from 104 participants were analyzed.

Sample composition (aMCI, n=64; AD with MMSE >15, n=40), size, and diagnostic criteria were based on a previous study (Reger, Watson et al. 2008). Forty participants (15 placebo, 13 low dose insulin and 12 high dose insulin) completed the PET sub-study, and 23 participants (n=8 placebo and 15 insulin) completed the LP sub-study. Diagnoses were determined by expert physician and neuropsychologist consensus. Participants, caregivers, and all personnel involved in data collection were blinded to treatment

Figure 1 | Trial Enrollment Flow



assignment. Groups did not differ in education, body mass index, MMSE, gender, diagnosis, cholinesterase inhibitor treatment, or apolipoprotein E (APOE) ε4 allele carriage (Table 1).

**Table 1 | Participant Characteristics** 

| | Placebo<br>(n=30) | Low Insulin<br>(n=36) | High Insulin<br>(n = 38) |
|---|---|---|---|
| Age (mean yrs, SEM) | 74.9 (1.6) | 72.8 (1.5) | 69.9 (1.4)* |
| Education (mean yrs, SEM) | 15.3 (0.6) | 15.5 (0.5) | 16.2 (0.5) |
| 3MSE (mean, SEM) | 84.2 (2.7) | 83.7 (2.5) | 84.3 (2.4) |
| BMI (mean kg/m <sup>2</sup> , SEM) | 27.4 (0.8) | 26.7 (0.8) | 26.9 (0.7) |
| Gender (%F/M) | 43.3%/56.7% | 38.9%/61.1% | 47.4%/52.6% |
| A ChEl Treatment (%No/Yes) | 60%/40% | 72.2%/27.8% | 65.8%/34.2% |
| APOE-s4 Carriers (%No/Yes) | 55.2%/44.8% | 50%/50% | 57.9%/42.1% |
| Diagnosis (%MCI/AD) | 70%/30% | 55.6%/44.4% | 60.5%/39.5% |

<sup>\*</sup>High dose<placebo, p<0.05

Participants in the high dose insulin group were younger than placebo-assigned participants (p=0.02), whereas no differences were observed between placebo and low dose insulin groups. Age was included as a covariate in all analyses.

#### 3.2 **Procedures**

Participants were randomized to receive 10 International Units INI bid for a total daily dose of 20 International Units INI (n=36), 20 International Units INI bid for a total dose of 40 International Units (n=38) or placebo (saline bid, n=30) for 4 months. Participants were stratified by APOE- $\epsilon$ 4 carriage. Saline or insulin (Novolin R, Novo) was administered after breakfast and dinner with ViaNase  $^{\text{TM}}$ , an intranasal delivery system (Craft, Baker et al. 2012). Parallel versions of the cognitive protocol were administered at baseline, and months 2 and 4 of treatment. Co-primary outcome measures were delayed story recall and the DSRS which had previously demonstrated beneficial effects of insulin (Reger, Watson et al. 2008). Secondary measures included the AD Assessment Scale for Cognition (ADAS-Cog) (Reger, Watson et al. 2008), a test comprised of measures of memory, orientation, and language, with higher scores reflecting impairment ranging from 0 (best) to 70 (worst), and the ADCS-Activities of Daily Living scale (ADCS-ADL) (Galasko, Bennett et al. 1997). Baseline and post-treatment fasting CSF was analyzed for A $\beta$ 42 and tau with multi-parameter bead-based immunoassay INNO-BIA AlzBio3 (Innogenetics NV). Resting PET images were obtained using a GE Advance PET scanner (GE Medical Systems, Milwaukee, WI) using a previously described protocol (Baker, Cross et al. 2011).

## 3.3 Safety and Compliance

Support persons supervised participants' intranasal administration. Blood glucose was measured daily for the first week and then weekly; no group changes were observed over the course of the study (Craft, Baker et al. 2012). Compliance was monitored by quantifying unused drug. Safety data were reviewed semi-annually by a Data and Safety Monitoring Board. Adverse event reporting followed standard guidelines.

## 3.4 Statistical Analyses

For the intent-to-treat (ITT) sample, co-primary (delayed story recall and DSRS) and secondary (ADAS-Cog and ADAS-ADL) scores were log transformed. Scores were first subjected to mixed model repeated ANCOVA including all treatment groups (placebo, low dose insulin or high dose insulin) as the between subjects factor, and time (baseline, month 2, month 4) as the repeated factor using the SAS v9.2 General Linear Models procedure. After a significant (p<0.05) time by treatment group interaction reflecting a different pattern of change, each of the two insulin groups was compared separately with the placebo group using repeated measures ANCOVAs. Effect sizes (Cohen's f2) were calculated for all significant effects. Age was included as a covariate in all analyses. Diagnosis (aMCI or AD), gender, APOE-ε4 carriage status (yes or no), baseline 3MSE score, and years of education were also included as covariates. Non-significant covariates were dropped from the model. Significant relationships with covariates were explored with Pearson correlation (continuous variables) or follow-up ANOVAs (class variables). Missing values were treated with multiple imputation (Rubin 1987). For exploratory CSF biomarker analyses, because only a subset of participants elected to undergo LP and no differences were observed between the two insulin dose arms, the groups were combined into a single insulin-treated group to maximize power. Biomarkers were analyzed with the repeated ANCOVA strategy described above and, due to the small sample size, exploratory Spearman correlations were conducted to examine relationships among changes in biomarkers and outcome measures. Only study completers underwent post-treatment FDG-PET. Pre and post treatment scans were co-registered within subject and anatomically standardized to Talairach and Tournoux stereotactic coordinates (Talairach and Tournoux 1988, Minoshima, Koeppe et al. 1994). Pixel intensity was normalized to pontine values (Minoshima, Frey et al. 1995). Interval regional CMRqlc changes within groups were assessed using voxel-wise one-sample t statistics (pre-/posttreatment pair) and probability integral conversion to z scores (Worsley, Evans et al. 1992). Interval changes in regional CMRglc were then compared between 1) low insulin vs. placebo groups, and 2) high insulin vs. placebo groups. Based on the number of voxels and smoothness of the statistical map, a Type I error rate was controlled at 0.05 to account for multiple comparisons (Worsley, Evans et al. 1992). The resulting statistical maps were visualized in three-dimensional stereotactic surface

projections.

## 3.5 Results: Cognitive and Functional Outcome Measures

The three groups did not differ at baseline on any outcome measure; change from baseline is represented in figures for ease of interpretation. A significant overall treatment group by time interaction was observed for primary outcome delayed story recall (p=0.005). Compared to placebo, the low dose group had improved delayed recall (Fig. 2A; treatment by time p=0.02. Cohen's f2=0.36), whereas no effect was observed for the high dose group. Exploratory post-hoc analyses were then conducted to more closely examine the relationship of insulin dose to story recall, as this was a primary goal of this pilot clinical trial. Given findings that delayed recall may not be a sensitive measure for AD subjects due to increased variability and floor effects (Sano, Raman et al. 2011) we constructed a total story recall score (immediate and delayed), which showed improvement for the high-dose group (time by treatment interaction p<0.05, mean log total story recall change score with SEM = -.15(.1) for placebo vs.12 (.09) for the high dose group). A significant overall treatment by time interaction was observed for the other primary outcome measure, the DSRS (p=0.008). Compared with placebo, DSRS scores were preserved for both low and high dose groups (Fig.2B; treatment by time ps=0.01 and 0.01, Cohen's f2=0.38 and 0.41). For secondary measures, significant effects were observed for the ADAS-Cog (overall treatment by time interaction p=0.004). Both low and high insulin groups had less decline in cognition compared with placebo (Fig. 2C; treatment by time ps=0.04 and p=0.002, Cohen's f2=0.27 and .40). Treatment effects on the ADAS-Cog interacted with age; for the high dose insulin group, greater improvement (lowered score) tended to be associated with younger age (r=.31, p=0.06). For the ADCS-ADL, no overall effects of treatment on daily function were observed. However, a significant interaction with diagnosis was observed for this measure (overall treatment by time by diagnosis interaction p=0.02). Participants with AD receiving either dose of insulin had preserved function compared with placebo-assigned participants with AD who showed slight decline, whereas participants with aMCI showed no change regardless of treatment assignment (interactions for the participants with AD in low and high dose groups compared with placebo, ps=0.01 and 0.02, Cohen's f=0.45 and 0.43; Fig. 2D). Adjustment for APOE-ε4 status, baseline MMSE score, cholinesterase inhibitor treatment, gender, and education did not affect the pattern of any result.

Figure 2 | Change (Month 4-baseline) in log scores for (A) delayed story recall, (B) DSRS, (C) ADAS-Cog and (D) ADCS-ADL.



#### 3.6 **Results: AD Biomarkers**

CSF A $\beta$ 42, A $\beta$ 40 and tau did not change for the placebo or insulin-treated groups as a whole. In exploratory analyses, however, for insulin-treated participants, increased CSF A $\beta$ 42 concentrations were associated with improved delayed story recall and ADCS-ADL scores, whereas decreased A $\beta$ 42 was associated with worse performance (Spearman rhos=.59, p=0.02 and .60, p=0.02). Similarly, decreased tau/A $\beta$ 42 ratios over the 4-month study period correlated with improved delayed story recall and better daily function on both ADAS-ADL and DSRS for insulin-treated participants (Spearman rhos=-.52, p=0.05, -.50, p=0.07, and .53, p=0.05). No significant correlations were observed for the placebo group.

## 3.7 Results: FDG-PET CMRglc

Compared with placebo-assigned participants, the lower dose insulin group showed reduced progression of hypometabolism in bilateral frontal, right temporal, bilateral occipital, and right precuneus and cuneus regions over the 4-month treatment period (Fig. 3 and Table 2). The higher dose insulin group showed even greater treatment effects (higher Z scores) indicating less hypometabolism progression in most regions and in left parietal cortex.

Figure 3 | Areas of hypometabolism at baseline (scan 1) and month 4 (scan 2), along with changes in hypometabolism (time 2-time 1) within each group and differences in change between placebo and low or high insulin groups (nasal insulin-placebo). Hotter floors indicate areas of greater hypometabolism from time 1 to time 2, and from placebo to insulin groups.



Table 2 | Z scores and stereotactic coordinates for areas of reduced progression for low and high does insulin groups compared to placebo

| | | Stere | o Coordi | nates |
|--------------------------------------|-----|-------|----------|-------|
| | Z | Х | У | Z |
| Low Dose Insulin - Placebo | | | | |
| Inferior occipital cortex (L) | 4.3 | 19 | -62 | -7 |
| Lateral temporo-occipital cortex (R) | 3.9 | -39 | -80 | 2 |
| Precuneus (R) | 3.8 | -3 | -73 | 23 |
| Superior temporal cortex (R) | 3.7 | -53 | -24 | 2 |
| Lateral occipital cortex (L) | 3.5 | 6 | -87 | 9 |
| Orbital frontal cortex | 3.2 | -1 | 48 | -16 |
| High Dose Insulin - Placebo | | | | |
| Orbital frontal cortex | 5.8 | 1 | 23 | -18 |
| Inferior occipital cortex (L) | 5.3 | 21 | -64 | -9 |
| Inferior parietal cortex (L) | 4.1 | 35 | -40 | 47 |
| Precuneus/Cuneus (R) | 4.1 | 3 | -80 | 18 |
| Lateral occipital cortex (L) | 3.7 | 26 | -85 | 11 |
| Medial fronto-parietal cortex (L) | 3.7 | 10 | -19 | 41 |
| Caudate (R) | 3.6 | -12 | 3 | 20 |

Positive value on the x coordinate indicates the left hemisphere.

Positive value on the y coordinate indicates anterior brain.

Positive value on the z coordinate indicates superior brain.

## 3.8 Safety and Compliance

No treatment-related serious adverse events (SAEs) occurred during the study; most adverse events (AEs) were minor, such as mild rhinitis. AEs with an occurrence of >5% in any group are listed in Table 3. The total AE mean was higher for the low dose group compared with placebo (low dose mean total AEs with standard error=1.44±0.20, placebo =0.80±.22, p=0.04), with a similar trend for the high dose and placebo group comparison (high dose mean total AEs =1.21±0.16, placebo =0.80±.22, p=0.10). Mean compliance (number of completed doses) ranged from 95-97% and did not differ across groups.

Table 3 | Total number of adverse events and percent of sample for all events occurring for at least 5% of the participants in any treatment group.

| | Placebo | Low Insulin | High Insulin |
|------------|----------|-------------|--------------|
| Total AEs | 27/56.7% | 55*172.2% | 51+/68.4% |
| Dizziness | 3/10% | 3/8.3% | 5/13.2% |
| Headache | 1/3.3% | 4/8.3% | 2/5.3% |
| Nose bleed | 0/0.0% | 6/8.3% | 3/2.6% |
| Rhinitis | 1/3.3% | 8/16.7% | 417.9% |
| URI | 2/6.7% | 2/5.6% | 1/2.6% |
| Fall | 2/6.7% | 1/2.8% | 1/2.6% |
| Rash | 2/6.7% | 1/2.8% | 2/2.6% |
| Other | 16/46.7% | 30/58.3% | 33/60.5% |

<sup>\*</sup> Low Insulin Total AEs > Placebo, p<0.05

## 3.9 **Implications**

These results suggest that adults with aMCI or AD may benefit from INI treatment. Compared with placebo, the lower dose of insulin improved delayed memory, and both insulin doses preserved caregiver-rated ability to carry out daily functions. General cognition as assessed with the ADAS-Cog, the primary outcome measure for the current trial, was also preserved by both doses of INI. In exploratory analyses, changes in CSF A $\beta$ 42 and tau/A $\beta$ 42 ratios were associated with cognitive and functional changes for insulin-treated participants. Placebo-assigned participants showed decreased CMRglc values in frontal, temporal, and parietal cortices as well as precuneus and cuneus over the 4-month period, whereas insulin-treated participants showed no decline. The longstanding FDG PET finding of posterior cingulate, precuneus and cuneus hypometabolism in AD has been hypothesized to be due to functional disconnection of the hippocampal formation, so enhanced metabolism and memory with INI may reflect enhanced hippocampal input to this region. Similarly there are strong connections between the posterior cingulate, precuneus, cuneus and prefrontal and superior temporal cortex (Cavanna and Trimble 2006), which may also be affected by INI. Finally, no treatment-related SAEs occurred. These promising results provide a strong rationale for the longer, larger, multi-site trial proposed in this application.

#### 4.0 **PRELIMINARY STUDY 2**

A follow-up study has recently concluded and results have been published (Craft et al. JAMA Neurology, 2020).

**Objectives:** This study tested the effects of 40 International Units of intranasal insulin administered daily for 12 months, compared with placebo, on cognition, daily function and safety in adults with MCI or mild AD. Longer-term effects were examined in a six-month open-label extension offered to all participants. Safety and feasibility issues relating to the use of intranasal delivery devices were also evaluated. The trial is nearing completion; all participants have concluded the blinded phase.

**Methods:** Twenty-six sites enrolled 289 participants with MCI or mild AD in this randomized, double-blind, Phase II/III trial (NCT01767909). Adults 45 to 85 years of age with diagnoses of amnestic MCI

<sup>+</sup>High Insulin Total AEs > Placebo, p<0.10

or AD (National Institute on Aging-Alzheimer's Association criteria) with Mini-Mental State Exam (MMSE) scores >19, Clinical Dementia Ratings (CDR) of 0.5 or 1, and delayed Logical Memory scores within a specified education-adjusted range were eligible. Participants with diabetes requiring medication were excluded, as were participants who had used insulin within one year of the screening visit. Participants were randomized on a 1:1 basis using a covariate-adaptive algorithm that weighted MMSE, apolipoprotein Ε-ε4 (APOE-ε4) allele carriage, study site, sex, and age based on previous work indicating these factors may impact treatment response. Participants received 40 International Units of insulin or insulin diluent placebo (Humulin R U-100 or insulin diluent, Eli Lilly, Indianapolis, USA) daily for 12 months. At the end of the 12-month blinded phase, all participants were offered open-label insulin treatment for 6 months. The primary outcome (Alzheimer's Disease Assessment Scale for Cognition-12/ADAS-Cog12) was administered at baseline and then at 3 month intervals. Secondary functional outcomes (Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale for MCI; CDR Sum of Boxes) were assessed at 6 month intervals, as was a memory composite (Free and Cued Selective Reminding Test and Story Recall). Cerebrospinal fluid biomarkers (Aβ42 and Aβ42/tau ratio) and magnetic resonance imaging hippocampal and entorhinal cortex volumes were measured at baseline and after 12 months.

Device issues. Intranasal delivery device monitoring revealed no safety issues. However, for the first 49 participants, the delivery device had frequent malfunctions (i.e. failure to turn on) that impacted dosing reliability. At that time, a newly available device was introduced (Precision Olfactory Device/POD, Impel NeuroPharma, Seattle, USA) which was used by the remaining 240 participants with good reliability.

**Results:** Demographic characteristics of enrolled participants are presented in Table 1. Retention was excellent, with only 25 participants discontinuing treatment during the blinded phase, and 15 also discontinuing study visits during the blinded phase. Quarterly DSMB reviews did not detect any safety issues and approved unmodified continuation of the trial.

Data from the subgroup of participants who used the POD were analyzed separately from the ViaNase group. The primary analysis of the POD group showed was negative; no difference in ADAS-Cog12 scores were observed after 12 months of INI treatment compared with placebo (Fig.1). In contrast, analysis of the ViaNase group showed beneficial effects of insulin compared with placebo; the effect was significant at 6 months (p<0.01), and persisted at 12 months (p=0.09; Fig. 2).

| Table 1. Baseline Participant | |
|-------------------------------|-----------------|
| Characteristics | |
| N (F/M) | 289 (134 / |
| | 155) |
| Age (years) | $70.95 \pm 7.1$ |
| Diagnosis | 105 / 184 |
| (MCI/AD) | |
| MMSE | $24.8 \pm 2.7$ |
| Logical | $2.1 \pm 2.7$ |
| Memory | |
| ΑΡΟΕ (ε4+/ε4- | 193 / 96 |
| ) | |





#### ADAS12 Mean Change from BL for ViaNase



Fig. 1 Fig. 2

**Implication:** These results suggest that the two delivery devices may be providing different doses of insulin to the CNS. The ViaNase device results are consistent with multiple previous studies. The POD had not been used previously in clinical trials with insulin, and thus was relatively untested in terms of delivery efficacy, although modeling in organoid nasal cavities was conducted to verify that the target amount of insulin was dispersed to the target location in the nasal cavity. These divergent results raise the possibility that specific characteristics of the device can affect delivery. Any future studies of intranasal insulin will need to utilize devices that have been demonstrated to effectively deliver insulin to the CNS. A study currently in progress compared delivery of two doses of insulin with 2 devices in order to provide supportive evidence for future trials.

#### 5.0 **PRELIMINARY STUDY 3**

**Objectives**: The Device Delivery Study compared whether delivery of 20 or 40 IU of insulin with the Aptar VP7 or CPS devices raised insulin acutely in CSF.

**Methods**: The study consists of a single site, randomized, double-blind trial comparing the acute effects of INI (20 or 40 International Units) delivered with the Aptar CPS or VP7 devices on CSF insulin levels, AD biomarkers and memory. At study entry, participants were randomized to the CPS or VP7 device. They were then randomized to receive either a 20 or 40 IU dose of insulin first, and the other dose on a second visit. Participants who were cognitively normal or who had aMCI (n=10) were enrolled. The primary outcome measure consisted of CSF insulin levels. Secondary measures included a memory test and CSF biomarker levels.

Two lumbar punctures were performed in the morning after a minimum 8-hour overnight fast at least a week apart. After insertion of the spinal catheter, blood and CSF was collected immediately. Insulin (20 or 40 IU) was then be administered, and additional CSF and blood was collected at 10 and 20 minutes following administration, after which the spinal catheter was withdrawn.

**Results**: Although the study is ongoing, preliminary analyses have been conducted to inform the design of the current trial. Change in CSF insulin from baseline values are shown below for individual participants (left) using the VP7 and CPS devices to administer 20 IU (Dose 1) and 40 IU (Dose 2). Mean change for the groups is shown on the right.





Results showed that the VP7 device did not reliably increase CSF insulin levels, with only one participant in the 40 IU dose showing elevations after administration. More reliable elevations were demonstrated with the CPS device, particularly for the 40 IU dose. All five participants showed increased CSF insulin after administration, and the average change was significant. Based on these

data, the CPS device has been selected for this pilot trial, as has the 40 IU dose.

## 5.1 Rationale for Dosage Selection

The dosage of insulin selected (40 International Units INI q.i.d.) has been used in multiple prior studies with positive results. The dosage of empa (10 mg q.d.) is also standard and has been used in previous large trials (EMPA-REG-OUTCOME).

#### 5.2 Rationale for Primary and Secondary Outcome Measures

Because no published study has examined the safety of empagliflozin in adults with Alzheimer's disease or in combination with intranasal insulin, the proposed study specifies safety, defined as number of treatment-related adverse events, as the primary outcome.

Regarding secondary measures, in previous studies intranasal insulin acutely improved cognitive performance and affected CSF levels of AD biomarkers as well as MRI measures of vascular integrity (Reger et al. 2008; Craft et al. 2012; Kellar et al. 2021). Thus examining effects on these measures will provide information to be used in the design of a future Phase II trial.

## 5.3 Rationale for Design of Trial

The proposed pilot study will provide safety and efficacy preliminary data regarding singular and combined effects of two therapeutic approaches, intranasal insulin and treatment with the SGLT2i empagliflozin, to correct bioenergetic and vascular dysfunction in adults with preclinical AD and amnestic mild cognitive impairment (aMCI) or early AD.

#### 5.4 Rationale for Biofluids

The CSF biomarkers insulin, A $\beta$ 42, A $\beta$ 40, total tau and phospho-tau will be measured, as well as CSF markers of vascular function. Plasma levels of insulin and glucose will be also assessed. Plasma and CSF samples obtained in this study will be banked so that other putative biomarkers may be measured by qualified investigators in the future given adequate rationale and feasibility.

#### 6.0 **STUDY OVERVIEW**

The study will consist of a single site, randomized, double-blind trial comparing the effects of 4 weeks of INI (40 International Units q.i.d.), empa (10 mg q.d.) and combined INI and empa compared with placebo on CSF biomarkers and cognition. At study entry, participants will be randomized to one of 4 conditions: INI, empa, INI+empa, placebo. Participants who are cognitively normal but have abnormal elevations of brain amyloid (n=20) or who have MCI or early AD (n=40) will be enrolled. The primary outcome measure will consist of safety (treatment-related serious adverse events). Secondary measures will consist of CSF biomarkers, cognition, and cerebral blood flow. Exploratory measures will include continuous glucose levels and sleep quality as assessed with actigraphy.

#### 6.1 **Study Population**

A total of 60 adults who are 1) cognitively normal/amyloid positive (n=20) or 2) diagnosed with aMCI or early AD (n=40) will be enrolled in this trial. To determine eligibility, all participants will undergo cognitive assessment, physical and neurological examination, ECG, clinical/safety laboratory assessment, and interviews of the participant and study partner conducted by the investigators and staff of the Clinical Core of the Wake Forest Alzheimer's Disease Research Center (ADRC).

## 6.2 **Diagnosis Criteria**

Diagnoses will be assigned by consensus of investigators from the Clinical Core of the Wake Forest ADRC using criteria specified by the NIA and Alzheimer's Association workgroups (Petersen, Doody et al. 2001, Albert, Dekosky et al. 2011).

Criteria for cognitively normal/amyloid positive adults:

- a) No evidence of significant cognitive impairment on objective testing
- b) Amyloid positivity as determined by amyloid PET (amyloid SUVR>1.21 or CSF A $\beta$ 42<600 pg/ml)

Diagnosis of aMCI or AD dementia requires:

- a) Diagnosis of amnestic mild cognitive impairment (MCI) or early AD according to NIA-Alzheimer's Association Criteria (CDR 0.5 or 1, MMSE>21)
- b) Amyloid positivity as determined by amyloid PET (amyloid SUVR>1.21 or CSF Aβ42<600 pg/ml)</li>

#### 6.3 **Inclusion Criteria**

The following inclusion criteria will be used:

- 1. Age 55 to 85 (inclusive)
- 2. Fluent in English
- 3. Cognitively normal or diagnosis of aMCI or mild AD
- 4. Amyloid positive by PET or CSF criteria
- 5. Stable medical condition for 3 months prior to screening visit
- 6. Stable medications for 4 weeks prior to the screening and study visits (exceptions may be made on a case by case basis by study physician)
- 7. Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be clinically insignificant by the study physician

## 6.4 Exclusion Criteria

The following exclusion criteria will be used:

- 1. A diagnosis of dementia other than AD
- 2. History of a clinically significant stroke
- Current evidence or history in past two years of epilepsy, head injury with loss of consciousness, any major psychiatric disorder including psychosis, major depression, bipolar disorder
- 4. Diabetes (type I or type II) insulin dependent and non-insulin dependent diabetes mellitus
- 5. Current or past regular use of insulin or any other anti-diabetic medication within 2 months of screening visit
- 6. History of seizure within past five years
- 7. Pregnancy or possible pregnancy
- 8. Use of anticoagulants, unless documentation received from prescribing clinician that anticoagulant medication can be held before LP, and approved by study clinician
- 9. Residence in a skilled nursing facility at screening
- 10. Use of an investigational agent within two months of screening visit

11. Regular use of alcohol, narcotics, anticonvulsants, anti-parkinsonian medications, or any other exclusionary medications (exceptions may be made on a case by case basis by study physician)

## 6.5 Recruitment and Retention Strategies

Recruitment will occur primarily from the Clinical Core of the Wake Forest ADRC. Some participants may also be identified from community recruitment efforts or from recently completed studies.

#### 7.0 **STUDY TIMELINE**

The approximate timeline for this 18-month study is projected as follows: 1) approximately two months for study startup activities; 2) study visits will occur over a ten-month period; 3) CSF and blood analyses, data analyses and study dissemination will occur over the final 6 months.

#### 8.0 **DESCRIPTION OF STUDY VISITS**

The "Schedule of Study Procedures and Assessments" in Table 4 (located in section 23.0) provides an overview of study visit activities. Genotyping will occur at Screening for participants who have not previously received APOE genotypes through the ADRC.

## 8.1 Screening (Visit 1)

The purpose of this visit is to determine study eligibility. Potential participants must sign an informed consent form and HIPAA Authorization prior to administration of any study-related procedures. After consent is obtained, participants will be given the MMSE, the CDR and Story Recall to determine study eligibility. Screening may be waived for participants who have received evaluations from the ADRC within the past 12 months. In addition, all cognitively normal participants must have amyloid PET or CSF  $A\beta42$  results available from the ADRC or affiliated studies prior to screening.

Information regarding demographics, concurrent medications, medical history and adverse events will be gathered from the participant. Vital signs, height and weight will be measured. A brief physical and neurological examination (which include a nasal examination) and a resting ECG will be performed. The ECG report will be reviewed, signed, and dated by the investigator or a medically qualified staff member as delegated by the Principal Investigator. Those with clinically significant ECG findings will be referred for follow-up as deemed appropriate by the investigator. These procedures may be waived for participants who have received evaluations from the ADRC within the past 12-months.

Fasting blood will be drawn for routine clinical laboratory evaluations. If values are outside of the laboratory's normal range and determined clinically significant by the medically qualified study investigators, lab tests may need to be repeated and may be considered exclusionary for participation in the study. Blood samples will also be collected for ApoE genotyping and DNA storage.

## 8.2 Baseline Visit 1 (Visit 2)

Results from all screening procedures must be reviewed and all inclusion/exclusion criteria must be met prior to proceeding to baseline. For participants whose screening visit was waived because they had received ADRC evaluations within the past 12-months will sign an informed consent form and HIPAA Authorization prior to administration of any study-related procedures.

According to the randomization schedule, the participant will be assigned to the insulin, empa, insulin+empa or placebo arm. On their first baseline visit they will receive the following:

- 1) Cognitive assessment
- 2) MRI (ADRC MRI may be used if done within 6 months of enrollment)
- 3) Insertion of the Libre Freestyle Pro continuous glucose monitor

- 4) Training on use of the Libre Freestyle Pro continuous glucose monitor
- 5) Training on how to use the intranasal delivery device and provision of saline to use with the device for the 1 week practice period (if applicable)
- 6) Training on how to record compliance
- 7) Training on use of the Empatica E4 actigraph for sleep assessment
- 8) PROMIS Sleep Disturbance and Sleep-Related Impairment Questionnaires
- 9) Patient Health Questionnaire-9 (PHQ-9)
- 10) General Anxiety Disorder Scale (GAD-7)
- 11) Nasal examination
- 12) Vital signs and weight
- 13) Collection of AEs and Con Meds

## 8.3 Baseline Visit 2 (Visit 3; one week after Baseline Visit 1)

For the 2<sup>nd</sup> baseline visit which occurs one week after Baseline Visit 1, the following procedures will be administered:

- 1) Lumbar puncture will be performed in the morning after a minimum 8-hour overnight fast. After insertion of the spinal catheter, CSF will be collected immediately. Insulin (40 IU) will then be administered, additional CSF will be collected following administration, and then the spinal catheter will be withdrawn. Blood will be drawn immediately before and following the LP under fasting conditions. Participants will then receive a snack and instructions about post-lumbar puncture care. Site staff will call the participant within 24 hours from the lumbar puncture procedure to inquire about the participant's well-being and possible adverse events.
- 2) The ADCS-ADL-MCI and gDRS will be administered
- 3) The Libre Freestyle Pro continuous glucose monitor will be removed
- 4) The Empatica E4 actigraph and PROMIS sleep questionnaires will be collected
- 5) Device use and feasibility issues during the run-in period will be reviewed
- 6) Distribution of study drug and placebos (if applicable)
- 7) Nasal examination
- 8) Vital signs and weight
- 9) Collection of AEs and Con Meds

# 8.4 Re-supply Visit and Safety/Compliance Assessment 1 (Visit 4; one week after Baseline Visit 2)

For the re-supply visit, the following procedures will be administered:

- 1) Device use and instructions will be reviewed
- 2) Collection of nasal drug vial and pill count
- 3) Distribution of study drug and placebos (if applicable)
- 4) Vital signs and weight
- 5) Collection of AEs and Con Meds

## 8.5 Phone Safety/Compliance Assessment 2

Participants will receive a call from study staff 2 weeks after initiating treatment to monitor for adverse events and compliance.

#### 8.6 **Post-treatment Visit 1 (Visit 5)**

On their first post-treatment visit they will receive the following:

- 1) Cognitive assessment
- 2) MRI
- 3) Insertion of the Libre Freestyle Pro continuous glucose monitor
- 4) Provision of the Empatica E4 actigraph for sleep assessment

- 5) PROMIS Sleep Disturbance Questionnaires
- 6) Patient Health Questionnaire-9 (PHQ-9)
- 7) General Anxiety Disorder Scale (GAD-7)
- 8) Nasal examination
- 9) Vital signs and weight
- 10) Collection of AEs and Con Meds

## 8.7 Post-treatment Visit 2 (Visit 6; one week after Post-treatment Visit 1)

On their second post-treatment visit which occurs 1 week after Post-treatment Visit 1 they will receive the following:

- 1) Lumbar puncture will be performed in the morning after a minimum 8-hour overnight fast. After insertion of the spinal catheter, CSF will be collected immediately. Insulin (40 IU) will then be administered, additional CSF will be collected following administration, and then the spinal catheter will be withdrawn. Blood will be drawn immediately before and following the LP under fasting conditions, including routine clinical laboratory evaluations. Participants will then receive a snack and instructions about post-lumbar puncture care. Site staff will call the participant within 24 hours from the lumbar puncture procedure to inquire about the participant's well-being and possible adverse events.
- 2) The ADCS-ADL-MCI and qDRS will be administered
- 3) The Libre Freestyle Pro continuous glucose monitor will be removed
- 4) The Empatica E4 actigraph and sleep questionnaire will be collected
- 5) Nasal examination
- 6) Vital signs and weight
- 7) Collection of AEs and Con Meds
- 8) Collection of nasal drug vials and pill count

Order of administration of procedures may occasionally vary due to scheduling constraints, as approved by the study clinicians.

## 9.0 STUDY-SPECIFIC PROCEDURES

#### 9.1 Cognitive Evaluation Instruments Administered to the Participant

Objective tests of cognitive function will include tests comprising the PACC5 (MMSE, Story Recall, the Rey Auditory Verbal Learning Test, Verbal Fluency), the CDR, and the ADAS-Cog14.

#### 9.2 Clinical and Functional Evaluations

## 9.2.1 Quick Dementia Rating System (QDRS)

The QDRS (Galvin, 2015) is a clinical scale that rates the severity of dementia as absent, questionable, mild, moderate, or severe (CDR score of 0, 0.5, 1, 2, or 3, respectively). The score assesses six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. At Screening the QDRS global score will be used for eligibility purposes. For all other administrations, the 6 domain scores will be summed to get the QDRS Sum of Boxes (SB) score.

#### 9.2.2 Activities of Daily Living Scale for MCI/ADL-MCI

The ADL-MCI is an activities of daily living questionnaire aimed at detecting functional decline. In a structured interview format, informants are queried as to whether participants attempted each item in the inventory during the prior 4 weeks and their level of performance. The ADL-MCI scale discriminates well between normal controls and patients with mild AD or MCI. It has good test-retest

reliability. The questions focus predominantly on instrumental activities of daily living scales (e.g. shopping, preparing meals, using household appliances, keeping appointments, reading).

9.2.3. PROMIS Sleep Disturbance and Sleep-Related Impairment Questionnaires (Short Form). These 8-item forms ask participants to rate quality of sleep on a 5-point scale.

#### 9.2.4 Patient Health Questionnaire-9 (PHQ-9).

This widely-used 9 item questionnaire assesses depression.

#### 9.2.5 General Anxiety Disorder Scale (GAD-7)

This widely-used 7-item questionnaire assesses anxiety.

#### 10.0 **STUDY METHODS**

## 10.1 Safety Assessments

At each study visit, all participants will undergo a nasal examination and any occurrence of adverse events will be reviewed and documented; concomitant medications will be recorded as well. In addition, 24 hours after the Lumbar Puncture, each study participant, or a person designated to speak for them will be contacted by phone to confirm the participant's well-being and queried about any new adverse events. All adverse events will be reported to the study MD for review.

## 10.2 Physical and Neurological Examination

A brief physical examination will be performed by a medically qualified professional at the screening visit. A review of the major body systems will be performed for example: skin, head/ears/eyes/nose/throat (HEENT), cardiovascular, pulmonary, abdomen, musculoskeletal, neurological, and gastrointestinal. Assessments of height (Screening visit only), weight, and vital signs (systolic and diastolic blood pressure, pulse, temperature, and respiration) are included. Neurological examination will include an assessment of cranial nerves, strength, coordination, reflexes, sensation, tremor and gait at every study visit. A nasal examination will also be performed. The examination will assess irritation or other abnormalities of the nares.

#### 10.3 Electrocardiogram (ECG)

A resting ECG will be performed at Screening visit. The ECG report will be reviewed, signed, and dated by the study clinician. Those with clinically significant ECG findings will be referred for follow-up as deemed appropriate by the investigator and may be excluded from the study.

#### 10.4 Clinical Laboratory Evaluations

All routine laboratory samples will be analyzed by Laboratory Corporation of America (Labcorp). Lab reports will be reviewed, signed and dated by the study clinician. If a value is outside of the laboratory's normal range, the clinician will indicate if it is clinically significant or not. If clinically significant, lab tests may need to be repeated and follow up with the participant's PCP should occur.

## 10.5 **Actigraphy**

The Empatica E4 device (<a href="https://www.empatica.com/en-eu/research/e4/">https://www.empatica.com/en-eu/research/e4/</a>) will be used to assess sleep quality. It uses an accelerometer to assess physical activity and heart rate variability from which a sleep quality index is calculated.

#### 10.6 Continuous Glucose Monitoring

The Abbott Freestyle Libre Pro is a continuous glucose monitor (CGM) system; a thin filament sensor the size of a quarter covered with a waterproof patch will be placed by a clinician or qualified study team member on the back of the participant's upper arm and worn for 7 days, then removed by the participant. The sensor records and uploads glucose data every 15 min. A report of average glucose

levels and number of hyperglycemic/hypoglycemic episodes can be linked to events such as meals, sleep, and activity. Participants will be assessed over a 1-week period.

#### 11.0 **BIOMARKER STUDIES**

#### 11.1 **CSF**

All CSF samples will be collected in the morning before breakfast and after an overnight fast. Participants who are taking anticoagulants cannot be enrolled unless documentation is received from the prescribing clinician that the anticoagulant medication can be held before the LP visits, and is approved by a study clinician. Based on clinician judgment and depending on the clinical indication, it may be suitable to discontinue participants from their anti-platelet agent (e.g., aspirin, Plavix, NSAIDs) for 5-7 days prior to lumbar puncture and until at least 24 hours after lumbar puncture. It is not required that participants be discontinued from their anti-platelet agent in order to screen and enroll in the study.

A minimal total volume of CSF (~25 ml) will be required for this study. To clear any blood from minor trauma associated with needle insertion, the first 1-2 mL of CSF are discarded (or more if needed). Collected CSF is aliquoted into sterile microtubes. Approximately 2ml of CSF or volume per local laboratory requirements will be sent at ambient temperature to the CRU laboratory for protein, glucose and cell count. CSF will be immediately frozen upright on dry ice for at least 20 minutes then stored at -70 until analysis.

CSF samples will be used to measure levels of insulin, A $\beta$ 42, A $\beta$ 40, total tau, and phospho-tau181. Assays will be performed by the Wake Forest ADRC Biomarker Service. CSF samples will also be frozen and stored for future analysis of putative biomarkers.

#### 11.2 Blood Collection at Lumbar Puncture Visits

All samples will be collected in the morning before breakfast and after a minimum 8-hour overnight fast. Blood samples (26 mL) will be collected before and after insulin administration. Blood will be processed for fasting plasma insulin and glucose. Additional blood for plasma and serum will be processed and banked.

#### 11.3 Genetic Samples, Storage and Future Use

DNA will be extracted from participant blood samples and will be analyzed for ApoE genotyping. ApoE genotyping will be used as a weighting factor for the minimization strategy during randomization. This will allow secondary analyses of data on the impact of the ApoE genotype on putative biomarkers of AD, clinical outcome measures, and adverse events. ApoE genotyping will be performed by Dr. Tim Howard under the auspices of the ADRC Biomarker service using established protocols.

#### 12.0 STATISTICAL PLAN

Statistical analyses will be conducted by the ADRC Biostatistics Core. To address the Primary Aim, number of treatment-related SAEs will be subjected to a repeated measures analysis of variance with group and time as the repeated measures. Secondary analyses will examine the effect of diagnostic status (cognitively normal vs. MCI/AD). Secondary analyses will also examine treatment-related differences for other CSF and plasma biomarkers, cognitive scores, and whole brain cerebral blood flow.

#### 12.1 **Power Analyses**

As this study is designed as a proof of concept study power calculations have not been conducted.

#### 13.0 **POTENTIAL RISKS**

## 13.1 Safety of Intranasal Insulin

Safety issues pertaining to INI administration for the treatment of diabetes have been extensively explored for over two decades (Pontiroli, Alberetto et al. 1982). For diabetes treatment, absorption enhancers must be used to increase the transport of insulin across the nasal membrane to the periphery due to the fact that peripheral bioavailablity of insulin without absorption enhancers is less than 1% (Illum 2002). A recent safety study of INI administration without absorption enhancers demonstrated no treatment induced changes in blood glucose levels, nasal airway patency, or transnasal pressure gradient (Kupila, Sipila et al. 2003). There are no known serious risks associated with INI without enhancers. A recent industry report raised the issue of rare but significant increases in lung cancer in smokers treated with inhaled insulin; six of 4740 patients taking inhaled insulin developed lung cancer compared with one of 4292 patients who received an active comparator (incidence per 100 patient years exposure, 0.13 vs 0.02). However, the inhaled insulin protocol used for diabetes treatment in this report included absorption enhancers to maximize delivery to lungs, whereas the nose-to-brain delivery device to be used in this study greatly minimizes lung delivery.

Regarding the risk of hypoglycemia, at least five peer reviewed human studies (Kern, Born et al. 1999, Born, Lange et al. 2002, Kupila, Sipila et al. 2003, Benedict, Hallschmid et al. 2004, Stockhorst, de Fries et al. Submitted for publication) and four preliminary studies (Reger, Watson et al. 2006, Reger, Watson et al. 2008, Reger, Watson et al. 2008) (Craft, Baker et al. 2012) revealed no change in blood glucose levels following intranasal insulin administration with doses that included 40 International Units 4 times daily for two months. There was one exception with the case of a single participant who experienced mild hypoglycemia (52 mg/dl) after skipping a meal and engaging in sustained vigorous exercise. In addition, a recent safety study (Kupila, Sipila et al. 2003) examined intranasal insulin administration of 60 International Units once a day for three weeks in 21 healthy adults. This randomized, double-blind, placebo-controlled crossover trial measured blood glucose levels six times a day during the first two and the last two days of treatment. Pre- and post-treatment blood laboratory tests and nasal examinations were performed. The nasal studies included rhinoscopy to detect local irritation, a saccharin particle test to analyze mucocilary clearance, and rhinomanometry to evaluate nasal airway patency and transnasal pressure gradient. Results indicated no change in blood glucose values with insulin, and no change in the frequency of glucose values above 3.0 mmol/L.

The only symptomatic hypoglycemic value occurred during placebo treatment. Insulin treatment had no effect on other laboratory values (C-peptide, total cholesterol, HDL, LDL, triglycerides, creatinine, glutamyl transferase), blood pressure, or body weight. In addition, nasal examinations revealed no adverse effects or functional disturbances following intranasal insulin administration. No serious adverse effects of treatment were observed in the preliminary studies (Reger, Watson et al. 2006, Reger, Watson et al. 2008, Reger, Watson et al. 2008, Craft, Baker et al. 2012).

#### 13.1 Safety of empagliflozin

SGLT2is including empagliflozin has been studied in multiple large trials of adults with Type 2 diabetes, as well as in non-diabetics with cardiovascular disease, and generally found to be safe (for a review, see Scheen, Nature, 2020). They are now considered standard of care for Type 2 diabetic patients with cardiovascular disease. Adverse effects that have been reported include: genital yeast infections especially in females, volume depletion, and diabetic ketoacidosis in the subset of Type 2 diabetic patients who have reduced insulin secretory capacity. Other effects may include frequent urination. Adults with seriously compromised kidney function (eGFR<45 mL/min/1.73m²) are not advised to take empa; kidney function will be assessed at the screening visit. Hypotension may also be observed rarely in patients with low systolic blood pressure, or who are taking diuretics. Participants will be monitored for hypotension and/or associate symptoms at each visit and during the two phone safety/compliance calls.

## 13.2 Safety of combined insulin and empagliflozin

Combined therapy of insulin and SGLT2is, including empa, was associated with rare but increased risk of ketoacidosis in the subset of Type 2 diabetic patients who have reduced insulin secretory capacity. Hypoglycemia has also been noted with combined administration, thought to be due to reduced hyperglycemia and related improvement in insulin sensitivity without concomitant reduction in insulin dosing. The proposed study will exclude participants with Type 2 diabetes, and will monitor blood glucose at all visits, as well as with continuous glucose monitoring during the last week of treatment. No other adverse interactions have been noted and SGLT2is are commonly prescribed for insulin-treated diabetics because of the multiple benefits on glycemic control and vascular function (Scheen, Nature, 2020).

#### 13.2 Risks associated with use of the Aptar CPS device

The Aptar CPS device has been extensively characterized and found to be safe for use. Participants could experience some discomfort to their eyes or face if they do not hold the device to their nose as directed; however, again, the study nurse will carefully instruct the participant regarding device use so that any errors can be immediately corrected.

- 13.3 Risks associate with use of the Empatica E4 actigraphy device Rarely, skin irritation may occur in reaction to the wristband or sensors.
- 13.4 Risks associated with use of the Libre Freestyle Pro Glucose Monitoring System The CGM is FDA-approved and widely used for assessing glucose levels in diabetes. The following are possible adverse effects of inserting a sensor and wearing the adhesive patch: local erythema (redness), local infection, inflammation, pain or discomfort, bleeding at the glucose sensor insertion site, bruising, itching, scarring or skin discoloration, hematoma, and adhesive irritation. There is a remote risk of sensor or needle fracture during insertion, wear or removal, with fragments retained under the skin.

#### 13.5 **Lumbar Puncture**

Lumbar puncture may be associated with pain during the performance of the procedure. This is usually temporary and confined to the lower back. Headache may occur in about 5% of elderly people who undergo lumbar puncture. Less commonly, in about 1-4% of participants, a persistent low-pressure headache may develop, probably due to leakage of CSF. Lower rates of post-LP headache have been noted in elderly patients, and when atraumatic (Sprotte) needles are used. If a post-LP headache persists it may need additional treatment, e.g. with fluids and analgesics. Uncommonly a blood patch (injection of some of the participant's blood to patch the CSF leak) may be needed. Potential but rare risks of lumbar puncture include infection, damage to nerves in the back, and bleeding into the CSF space. The risk of these is much less than 1%.

#### 13.6 **Blood Draw**

The risks of blood draw include pain from the needle, bruising or infection at the site of venipuncture, or fainting as a response to blood draw. Approximately 100 mLs of blood will be drawn for routine and biomarker laboratory assessments over the course of this study.

#### 14.0 PERSONNEL REQUIREMENTS

The following staff-member roles will be required to conduct the protocol.

Principal Investigator: The Principal Investigator (PI; Suzanne Craft, PhD) is responsible for the
overall conduct of the study. The PI will perform or supervise clinical evaluation of all participants
and ensure protocol adherence. The PI will supervise project personnel and ensure that clinical
raters maintain a high level of skill and accuracy in conducting assessments.

- Study Physicians: Don McClain, MD, PhD and James Tray Bateman, MD, MHS will serve as Study Physicians for the trial. Dr. McClain is a diabetologist with extensive experience in prescribing and monitoring SGLT2is and review all safety data for the trial as well as provide consultation as needed. Dr. Bateman is a Behavioral Neurologist with extensive experience in the assessment and care of older adults with Alzheimer's disease. He will be responsible for conducting and supervising the medical evaluation (nasal examination, physical and neurological examinations), reviewing adverse events, interpreting laboratory results, and supervising clinical care provided to the participant during the study. He will also supervise, and on some occasions may perform the lumbar punctures.
- **Study Clinician:** Samantha Rogers, PA-C, will conduct the majority of the lumbar punctures. She has conducted more than 300 lumbar punctures for the ADRC and affiliated studies over the past 5 years.
- Study Nurse/Coordinator: Deborah Dahl, RN will serve as Study Nurse/Coordinator for the trial. She will be responsible for managing the day-to-day conduct of the trial. Duties may include tracking recruitment, ensuring accurate administration of all instruments at the site, maintaining case report forms, processing of laboratory samples, and coordinating clinic visits. She will also oversee the use and maintenance of the devices, and coordinate with the Pharmacy regarding ordering and storage of saline and insulin.
- Interviewer/Psychometrician: This person will be responsible for administering the memory assessments.
- QDRS Rater: This person will render the QDRS rating based on clinical assessment of participant and study participant.
- Regulatory Affairs: Sarah Bohlman, MSL will be responsible for managing all regulatory related documents for the duration of the trial.

#### 15.0 **STUDY DRUGS**

Participants will take empa or placebo 30 minutes before breakfast daily. Participants will also take four doses of INI (40 International Units per dose) or placebo 30 minutes before each meal and 30 minutes before bedtime.

#### 15.1 Humulin® R U-100 Insulin

Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company) is a polypeptide hormone structurally identical to human insulin synthesized through rDNA technology in a special non-disease-producing laboratory strain of *Escherichia coli* bacteria. Humulin R U-100 has the empirical formula  $C_{257}H_{383}N_{65}O_{77}S_6$  and a molecular weight of 5808 Da. Humulin R U-100 is a sterile, clear, aqueous, and colorless solution that contains human insulin (rDNA origin) 100 units/mL, glycerin 16 mg/mL and metacresol 2.5 mg/mL, endogenous zinc (approximately 0.015 mg/100 units) and water for injection. The pH is 7.0 to 7.8. Sodium hydroxide and/or hydrochloric acid may be added during manufacture to adjust the pH.

More information about the Humulin<sup>®</sup> R U-100 insulin, including risks, contraindication and adverse reactions can be found in the US package insert (USPI).

#### 15.2 Empagliflozin

Empagliflozin (Jardiance, Boehringer-Ingelheim) is a sodium glucose co-transporter2 inhibitor. The chemical name of empagliflozin is D-Glucitol,1,5-anhydro-1-C-[4-chloro-3-[[4-[[(3S)-tetrahydro-3-furanyl]oxy]phenyl]methyl]phenyl]-, (1S). Its molecular formula is C23H27CIO7 and the molecular weight is 450.91. Empagliflozin is a white to yellowish, non-hygroscopic powder. It is very slightly soluble in water, sparingly soluble in methanol, slightly soluble in ethanol and acetonitrile; soluble in 50% acetonitrile/water; and practically insoluble in toluene. Each film-coated tablet of JARDIANCE

contains 10 mg empagliflozin (free base) and the following inactive ingredients: lactose monohydrate, microcrystalline cellulose, hydroxypropyl cellulose, croscarmellose sodium, colloidal silicon dioxide and magnesium stearate. In addition, the film coating contains the following inactive ingredients: hypromellose, titanium dioxide, talc, polyethylene glycol, and yellow ferric oxide.

More information about empagliflozin can be found the prescribing information included on the Jardiance/Boehringer-Ingelheim website:

https://docs.boehringeringelheim.com/Prescribing%20Information/PIs/Jardiance/jardiance.pdf

#### 15.2 Randomization

Eligible participants will be randomized on a 1:1 schedule to placebo (insulin diluent; placebo capsule), INI, empa, or INI+empa. Randomization will be stratified by diagnosis (normal, MCI or AD)

## 15.3 **Blinding**

Neither participants nor site personnel involved in assessing participants will know which dose of insulin is being administered. Exceptions will be the study nurse who is directly involved in preparing the insulin.

## 15.4 **Study Drug Dispensing**

Study drug will be dispensed by the study nurse.

#### 15.5 **Intranasal Administration**

Insulin will be administered with the Aptar CPS delivery device. This device release a metered insulin dose into the participant's nose, allowing the administration of smaller particle sizes to increase deposition in the upper nasal cavity while minimizing transport to the lungs. A volume of about 0.7 mL of insulin will be administered in each nostril, for a total volume of 1.4 mL per dose, 4 times daily.

#### 15.6 **Storage**

Insulin and empa will be maintained at a controlled temperature.

#### 15.7 **Drug Accountability**

The study nurse coordinator will maintain a log of study drug usage.

#### 16.0 ADVERSE EVENTS

## 16.1 **Definition**

An adverse event (AE) is defined as per the Code of Federal Regulation Title 21 Part 312.

http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/cfrsearch.cfm?fr=312.32

Adverse events which occur after informed consent is signed include but are not limited to: (1) worsening or change in nature, severity, or frequency of conditions or symptoms present at the start of the study; (2) participant deterioration due to primary illness; (3) intercurrent illness; and (4) drug interaction. An abnormal laboratory value will only be reported as an AE if the investigator considers it to be an AE, or if it leads to the participant being withdrawn from the study.

The investigator should attempt to establish a diagnosis of the event based on signs, symptoms, and or other clinical information. In such cases, the diagnosis should be documented as the AE and not the individual signs or symptoms. Symptoms and conditions present at the beginning of the study will be characterized, so that AEs can be defined as any new symptom, or any increase in frequency or severity of an existing symptom.

Following questioning and evaluation, all AEs, whether determined to be related or unrelated to the study drug by a medically qualified site PI or clinician (MD, DO, NP or PA), must be documented in the participant's medical records, in accordance with the investigator's normal clinical practice, and on the AE *e*-CRF. Each AE is evaluated for duration, severity, seriousness, and causal relationship to the study drug.

## 16.2 **Following Up on AEs**

The investigator is obliged to follow participants with AEs until the events have subsided, the conditions are considered medically stable, or the participants are no longer available for follow up. Participants who discontinue due to adverse experiences will be treated and followed according to established medical practice. Adverse events will be rated as mild, moderate or severe. This will also pertain to abnormal laboratory values deemed clinically significant by the site clinician.

## 17.0 SERIOUS ADVERSE EVENTS (SAE)

#### 17.1 **Definition**

A serious adverse event is defined as per the Code of Federal Regulation Title 21 Part 312

http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/cfrsearch.cfm?fr=312.32

## 17.2 **Reporting SAEs**

Any serious and adverse event due to any cause, which occurs during the course of the investigation (i.e. any time after informed consent, regardless of study drug exposure), will be reported to the PI and study physician within 24 hours of learning of the event. All serious adverse events will be reported to the Wake Forest IRB within 7 days of study personnel learning of the event.

## 17.3 **IND Safety Reporting**

As the Sponsor of the IND related to this study, any unexpected fatal or life-threatening suspected adverse reactions will be reported to the FDA no later than 7 calendar days after the initial receipt of the information per 21 CFR 312.32(c)(2).

Reporting of any (1) serious, unexpected suspected adverse reactions (2) findings from other clinical, animal, or in-vitro studies that suggest significant human risk, and (3) a clinically important increase in the rate of a serious suspected adverse reaction no later than 15 calendar days after determining that the information gualifies for reporting per 21 CFR 312.32(c)(1).

#### 18.0 ETHICS & REGULATORY CONSIDERATIONS

#### 18.1 **Ethical Standard**

Study investigators are charged with conducting this study in full conformity with:

- 1. Good Clinical Practice (GCP) guidelines, as defined by the International Conference on Harmonisation (ICH) Guideline, Topic E6
- 2. The United States Code of Federal Regulations, Title 21, Part 50 (21CFR50) Protection of Human Subjects
- 3. 21CFR56 Institutional Review Boards (IRBs)
- 4. HIPAA
- 5. State and Federal regulations and all other applicable local regulatory requirements and laws.

Study personnel involved in conducting this study will be qualified by education, training and experience to perform their respective task(s) in accordance with GCP.

## 18.2 Institutional Review Board (IRB)

This protocol and the associated informed consent documents and recruitment material will be approved by the Wake Forest IRB which is registered with the Office for Human Research Protections (OHRP). Any amendments to the protocol or consent materials must also be approved before they are placed into use. The investigator shall notify the IRB of deviations from the protocol or serious adverse events occurring at the site, in accordance with local procedures.

#### 18.3 Informed Consent & HIPAA Authorization

In obtaining and documenting informed consent, the investigator should comply with the applicable regulatory requirement(s), and should adhere to GCP and to the ethical principles that have their origin in the Declaration of Helsinki. Prior to the beginning of the trial, the investigator should have the IRB's written approval of the written informed consent form (ICF) and any other written information to be provided to participants. Participants, their relatives, guardians, or authorized representatives and study partners will be given ample opportunity to inquire about the details of the study. Prior to a subject's participation in the trial, the written informed consent form and HIPAA Authorization should be signed and personally dated by the subject and/or the subject's legally authorized representative, the study partner and by the person who conducted the informed consent discussion. Participants should be provided a copy of the signed ICF.

The informed consent will not only cover consent for the trial itself, but for the genetic research, biomarker studies and biological sample storage. The consent for storage will include consent to access stored data and biological samples for secondary analyses. Consent forms will specify that DNA and biomarker samples are for research purposes only; the tests on the DNA and biomarker samples are not diagnostic in nature and participants will never receive results.

## 18.4 Participant Confidentiality | HIPAA

Participant confidentiality is strictly held in trust by the participating investigators, research staff, and the sponsoring institution and their agents. This confidentiality is extended to cover testing of biological samples and genetic tests in addition to the clinical information relating to participants. The study protocol, documentation, data and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party, without prior written approval. Any data, specimens, forms, reports, and other records that leave the site will be identified only by a subject identification number to maintain confidentiality. All records will be kept in a locked file cabinet. All computer entry and networking programs will be done using subject IDs only. Information will not be released without written permission of the subject, except as necessary for monitoring by the IRB, FDA, NIA, and the OHRP.

Information about subjects will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Those regulations require a signed HIPAA Authorization informing the subject of the following:

- What protected health information (PHI) will be collected from participants in this study
- Who will have access to that information and why
- Who will use or disclose that information
- The rights of a research participant to revoke their authorization for use of their PHI.

In the event that a subject revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information collected prior to the revocation of subject authorization. Each site PI, under the guidance of his/her IRB, is responsible for ensuring that all applicable HIPAA regulations and State laws are met.

#### 19.0 GENETIC RESEARCH & STORAGE OF GENETIC MATERIAL

The DNA is banked in locked freezers in the ADRC Biomarker Service. Sample tubes are bar-coded and linked to participant ID number only and banked without personal identifiers.

Only DNA from consenting participants will be banked and used to facilitate future research on aging and dementia, particularly in the discovery of genetic polymorphisms that may influence risk of developing AD. Collection of DNA will permit investigators to probe candidate genetic polymorphisms as predictors of outcome in future studies. The samples will be stored by the ADRC.

## 19.1 Storage of Biospecimen Samples

All biospecimens being banked for future AD biomarker research will be stored by the ADRC Biomarker Service. Participant will be asked to consent to allow samples to be used for future research.

#### 20.0 RISKS AND BENEFITS ASSOCIATED WITH THIS STUDY

## 20.1 Potential Benefits of the Proposed Research to Human Subjects

There is an urgent need to identify promising treatments for patients with AD and its prodrome aMCI. In a previous trial (Craft, Baker et al. 2012), intranasal insulin safely improved delayed memory and function in these patients. In a recent trial, these results were replicated with the subgroup of participants who used the ViaNase device, but not with the POD cohort. The proposed trial is designed to answer the important question of whether the Aptar CPS device is effective in delivering intranasal insulin into the CNS. This knowledge will enable the conduct of future Phase III trials of intranasal insulin.

There are no significant potential clinical benefits for the participants in this study. Rather, there is a clear scientific benefit for the field as a whole. The relatively minor risks posed by the intranasal administration, cognitive testing, and LP are outweighed by the value of the scientific investigations outlined in this study.

#### 20.2 Inclusion of Women and Minorities

There are currently no studies that definitively support or negate the existence of significant differences in response to intranasal insulin in subgroups defined by gender or ethnic background. A specific goal percentage for women and minority enrollment is not set for this study. However, we will monitor minority enrollment throughout the study and make special effort to encourage minority enrollment. Minority enrollment will be facilitated through minority outreach effort coordinated by the Recruitment Core at the ADRC. No participant will be excluded due to his or her sex, race, or ethnic group.

# 20.3 Inclusion of Children as Participants in Research Involving Human Subjects Children will not be included.

## 20.4 Data and Safety Monitoring Plan

The principal investigator and study clinician(s) will be responsible for the overall monitoring of the data and safety of study participants, with assistance by members of the study staff. Participants will be screened at the beginning of the study and will be monitored carefully at each study visit. Participants will be queried for serious adverse events (SAEs) and selected AEs (those temporally related to study procedures) at each study visit. All SAEs and selected AEs will be recorded on an AE case report form. Based on the nature of the AE, study clinicians will determine the severity of the event and association with the study. All serious adverse events will be reported. Serious adverse events are defined as events that are (1) life-threatening or fatal, (2) result in severe or permanent disability, or (3) require hospitalization. SAEs will be reported to the IRB within 7 days of investigator

knowledge of the event if they are related and unanticipated (i.e. if they qualify as an unanticipated problem). All serious adverse events will be followed until resolution, or 90 days after study participation has been terminated.

"Severity" of events will be graded according to the following guidelines:

- 1. Mild: The participant is aware of, but can easily tolerate, the event
- 2. Moderate: The discomfort of the event is severe enough to interfere with some usual activities
- 3. Severe: The participant is incapacitated, and unable to perform most or all usual activities

The "study-relatedness" will be assigned according to the following guidelines:

- 1. Definitely Related: The reaction follows a reasonable temporal sequence and is known to be an effect of participation or a procedure
- 2. Possibly Related: The reaction follows a reasonable temporal sequence, and current medical knowledge does not preclude a relationship between participation or procedure and the event.
- 3. Unlikely: Little evidence to suggest a causal relationship (e.g. the event did not occur within a reasonable time after administration of the trial medication) or another reasonable explanation for the event (e.g. another clinical condition or other concomitant treatment).
- 4. Definitely Unrelated: Current medical knowledge precludes a causal relationship between participation or procedure and the event or the cause of the reaction is known to be other than participation or procedure.

#### 21.0 PUBLICATION POLICY

The results of this study may be published, depending on the results.

#### 22.0 SHARING OF FINAL RESEARCH DATA

Data from this research will be shared with other researchers pursuant to the 02/26/2003 "NIH Final Statement on Sharing Research Data". NIH believes that data sharing is important for further translation of research results into knowledge, products, and procedures to improve human health. The NIH endorses the sharing of final research data to serve these and other important scientific goals. To protect subjects' rights and confidentiality, identifiers will be removed from the data before they are shared.

# 23.0 TABLE 4: SCHEDULE OF PROCEDURES AND ASSESSMENTS

| Visit # | 1 | 2 | 3 | 4 | | 5 | 6 |
|---|---|---|---|---|---|---|---|
| Visit Name | Screen <sup>2</sup> | Baseline<br>V1 | Baseline<br>V2 | Re-<br>supply | Phone | Post-<br>Treatment<br>V1 | Post-<br>Treatment<br>V2 |
| 1.6 | | | | | | | |
| Informed<br>Consent | X | X <sup>3</sup> | | | | | |
| Demographics | Χ | X <sup>3</sup> | | | | | |
| Medical History | X | X <sup>3</sup> | | | | | |
| Concomitant<br>Meds | X | X | Х | X | Х | Х | X |
| Adverse Events | X | X | X | Χ | Χ | X | X |
| Nasal Exam | Χ | Х | X | | | X | X |
| Physical and<br>Neurological<br>Exam | X | | | | | | |
| Vital Signs | Х | Х | Х | Χ | | X | Х |
| Height | Х | | | | | | |
| Weight | Χ | Х | Х | Х | | Х | Х |
| ECG | Х | | | | | | |
| Cognitive<br>Assessment | Х | Х | Х | | | Х | Х |
| Questionnaires | Х | Х | Х | | | X | Х |
| Aptar CPS Device & Compliance Training | | Х | | | | | |
| Compliance<br>Assessment | | | Х | X | X | X | X |
| Study Drug<br>Dispensed | | | X <sup>4</sup> | Х | | | |
| Actigraphy | | Х | | | | Х | |
| Continuous Glucose Monitor (CGM) Placement | | Х | | | | Х | |
| Blood Draw | Χ | | Х | | | | Х |
| - Clinical<br>Labs | Х | | Х | | | | Х |
| - ApoE<br>Genotyping<br> DNA<br>Banking | Х | | | | | | |
| - Biomarkers<br> Plasma <br>Serum <br>Sample<br>Banking | | | Х | | | | X |
| LP | | | Х | | | | Х |

| - CSF<br>Biomarkers<br> Banking | | Х | | х |
|---|---|---|---|---|
| - Post-<br>Procedure<br>Safety<br>Telephone<br>Check | | X | | Х |
| MRI | X <sup>1</sup> | | Х | |

<sup>&</sup>lt;sup>1</sup>MRI can be excluded if done within 6 months of enrollment

<sup>&</sup>lt;sup>2</sup>Screening may be waived if evaluations have been performed within the last 12 months <sup>3</sup>Will be performed if participant was eligible to skip Screening

<sup>&</sup>lt;sup>4</sup>Study drug may be re-dispensed as needed (if applicable)

- Albert, M. S., S. T. Dekosky, D. Dickson, B. Dubois, H. H. Feldman, N. C. Fox, A. Gamst, D. M. Holtzman, W. J. Jagust, R. C. Petersen, P. J. Snyder, M. C. Carrillo, B. Thies and C. H. Phelps (2011). "The diagnosis of mild cognitive impairment due to Alzheimer's disease: Recommendations from the National Institute on Aging and Alzheimer's Association workgroup." <u>Alzheimers Dement</u>. Baker, H. and R. F. Spencer (1986). "Transneuronal transport of peroxidase-conjugated wheat germ agglutinin (WGA-HRP) from the olfactory epithelium to the brain of the adult rat." <u>Exp Brain Res</u> **63**(3): 461-473.
- Baker, L. D., D. J. Cross, S. Minoshima, D. Belongia, G. S. Watson and S. Craft (2011). "Insulin resistance and Alzheimer-like reductions in regional cerebral glucose metabolism for cognitively normal adults with prediabetes or early type 2 diabetes." <u>Arch Neurol</u> **68**(1): 51-57.
- Balin, B. J., R. D. Broadwell, M. Salcman and M. el-Kalliny (1986). "Avenues for entry of peripherally administered protein to the central nervous system in mouse, rat, and squirrel monkey." <u>J Comp Neurol</u> **251**(2): 260-280.
- Benedict, C., M. Hallschmid, A. Hatke, B. Schultes, H. L. Fehm, J. Born and W. Kern (2004). "Intranasal insulin improves memory in humans." <u>Psychoneuroendocrinology</u> **29**(10): 1326-1334. Benedict, C., W. Kern, B. Schultes, J. Born and M. Hallschmid (2008). "Differential sensitivity of men and women to anorexigenic and memory-improving effects of intranasal insulin." <u>J Clin Endocrinol Metab</u> **93**(4): 1339-1344.
- Bodian, D. and H. A. Howe (1941). "Experimental studies on intraneuronal spread of poliomyelitis virus." <u>Bull Johns Hopkins Hosp</u> **68**: 248-267.
- Born, J., T. Lange, W. Kern, G. P. McGregor, U. Bickel and H. L. Fehm (2002). "Sniffing neuropeptides: a transnasal approach to the human brain." Nat Neurosci **5**(6): 514-516.
- Broadwell, R. D. and B. J. Balin (1985). "Endocytic and exocytic pathways of the neuronal secretory process and trans-synaptic transfer of wheat germ agglutinin-horseradish peroxidase in vivo." <u>J Comp</u> Neurol **242**(4): 632-650.
- Cavanna, A. E. and M. R. Trimble (2006). "The precuneus: a review of its functional anatomy and behavioural correlates." <u>Brain</u> **129**(Pt 3): 564-583.
- Chiu, S. L., C. M. Chen and H. T. Cline (2008). "Insulin receptor signaling regulates synapse number, dendritic plasticity, and circuit function in vivo." Neuron **58**(5): 708-719.
- Craft, S., L. D. Baker, T. J. Montine, S. Minoshima, G. S. Watson, A. Claxton, M. Arbuckle, M. Callaghan, E. Tsai, S. R. Plymate, P. S. Green, J. Leverenz, D. Cross and B. Gerton (2012). "Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial." <u>Arch Neurol</u> **69**(1): 29-38.
- Craft, S., L. D. Baker, T. J. Montine, S. Minoshima, G. S. Watson, A. Claxton, M. Arbuckle, M. Callaghan, E. Tsai, S. R. Plymate, P. S. Green, J. Leverenz, D. J. Cross and B. Gerton (2012). "Intranasal Insulin Therapy for AD and MCI: A Pilot Clinical Trial." Arch Neurol **69**: 29-38.
- Craft, S., E. Peskind, M. W. Schwartz, G. D. Schellenberg, M. Raskind and D. Porte, Jr. (1998). "Cerebrospinal fluid and plasma insulin levels in Alzheimer's disease: relationship to severity of dementia and apolipoprotein E genotype." <u>Neurology</u> **50**(1): 164-168.
- Craft S, Raman R, Chow TW, Rafii MS, Sun CK, Rissman RA, Donohue MC, Brewer JB, Jenkins C, Harless K, Gessert D, Aisen PS. Safety, Efficacy, and Feasibility of Intranasal Insulin for the Treatment of Mild Cognitive Impairment and Alzheimer Disease Dementia: A Randomized Clinical Trial. JAMA Neurol. 2020 Sep 1;77(9):1099-1109. doi: 10.1001/jamaneurol.2020.1840. PMID: 32568367; PMCID: PMC7309571.
- Craft, S. and G. S. Watson (2004). "Insulin and neurodegenerative disease: shared and specific mechanisms." Lancet Neurol **3**(3): 169-178.
- De Felice, F. G., M. N. Vieira, T. R. Bomfim, H. Decker, P. T. Velasco, M. P. Lambert, K. L. Viola, W. Q. Zhao, S. T. Ferreira and W. L. Klein (2009). "Protection of synapses against Alzheimer's-linked toxins: insulin signaling prevents the pathogenic binding of Abeta oligomers." <u>Proc Natl Acad Sci U S A 106</u>(6): 1971-1976.

- Faber, H. K. (1938). "The early lesions of poliomyelitis after intranasal inoculation." <u>J Pediat</u> **13**(1): 10-37
- Fairbrother, R. W. and E. W. Hurst (1930). "The pathogenesis of, and propagation of the virus in, experimental poliomyelitis." J Path Bact **33**: 17-45.
- Fishel MA, Watson GS, Montine TJ, Wang Q, Green PS, Kulstad JJ, Cook DG, Peskind ER, Baker LD, Goldgaber D, Nie W, Asthana S, Plymate SR, Schwartz MW, Craft S.
- Arch Neurol. 2005 Oct;62(10):1539-44. "Hyperinsulinemia provokes synchronous increases in central inflammation and beta-amyloid in normal adults."
- Francis, G. J., J. A. Martinez, W. Q. Liu, K. Xu, A. Ayer, J. Fine, U. I. Tuor, G. Glazner, L. R. Hanson, W. H. Frey, 2nd and C. Toth (2008). "Intranasal insulin prevents cognitive decline, cerebral atrophy and white matter changes in murine type I diabetic encephalopathy." <u>Brain</u> **131**(Pt 12): 3311-3334. Frey, W. H. (2002). "Intranasal delivery: Bypassing the blood-brain barrier to deliver therapeutic

agents to the brain and spinal cord." Drug Delivery Technology 2(5): 46-49.

- Frolich, L., D. Blum-Degen, H. G. Bernstein, S. Engelsberger, J. Humrich, S. Laufer, D. Muschner, A. Thalheimer, A. Turk, S. Hoyer, R. Zochling, K. W. Boissl, K. Jellinger and P. Riederer (1998). "Brain insulin and insulin receptors in aging and sporadic Alzheimer's disease." <u>J Neural Transm</u> **105**(4-5): 423-438.
- Galasko, D., D. Bennett, M. Sano, C. Ernesto, R. Thomas, M. Grundman and S. Ferris (1997). "An inventory to assess activities of daily living for clinical trials in Alzheimer's disease. The Alzheimer's Disease Cooperative Study." <u>Alzheimer Dis Assoc Disord</u> **11 Suppl 2**: S33-39.
- Gasparini, L., G. K. Gouras, R. Wang, R. S. Gross, M. F. Beal, P. Greengard and H. Xu (2001). "Stimulation of beta-amyloid precursor protein trafficking by insulin reduces intraneuronal beta-amyloid and requires mitogen-activated protein kinase signaling." <u>J Neurosci</u> **21**(8): 2561-2570. Gil-Bea, F. J., M. Solas, A. Solomon, C. Mugueta, B. Winblad, M. Kivipelto, M. J. Ramirez and A. Cedazo-Minguez (2010). "Insulin levels are decreased in the cerebrospinal fluid of women with prodomal Alzheimer's disease." <u>J Alzheimers Dis</u> **22**(2): 405-413.
- Grillo, C. A., G. G. Piroli, R. M. Hendry and L. P. Reagan (2009). "Insulin-stimulated translocation of GLUT4 to the plasma membrane in rat hippocampus is PI3-kinase dependent." <u>Brain Res</u> **1296**: 35-45.
- Hallschmid, M., C. Benedict, B. Schultes, J. Born and W. Kern (2008). "Obese men respond to cognitive but not to catabolic brain insulin signaling." Int J Obes (Lond) **32**(2): 275-282.
- Hong, M. and V. M. Lee (1997). "Insulin and insulin-like growth factor-1 regulate tau phosphorylation in cultured human neurons." J Biol Chem **272**(31): 19547-19553.
- Hughes, C. P., L. Berg, W. L. Danziger, L. A. Coben and R. L. Martin (1982). "A new clinical scale for the staging of dementia." <u>Br J Psychiatry</u> **140**: 566-572.
- Illum, L. (2002). "Nasal drug delivery: new developments and strategies." <u>Drug Discov Today</u> **7**(23): 1184-1189.
- Kern, W., J. Born, H. Schreiber and H. L. Fehm (1999). "Central nervous system effects of intranasally administered insulin during euglycemia in men." Diabetes **48**(3): 557-563.
- Kristensson, K. and Y. Olsson (1971). "Uptake of exogenous proteins in mouse olfactory cells." <u>Acta Neuropathol</u> **19**(2): 145-154.
- Kupila, A., J. Sipila, P. Keskinen, T. Simell, M. Knip, K. Pulkki and O. Simell (2003). "Intranasally administered insulin intended for prevention of type 1 diabetes--a safety study in healthy adults." <u>Diabetes Metab Res Rev</u> **19**(5): 415-420.
- Lee, C. C., Y. M. Kuo, C. C. Huang and K. S. Hsu (2009). "Insulin rescues amyloid beta-induced impairment of hippocampal long-term potentiation." <u>Neurobiol Aging</u> **30**(3): 377-387.
- Minoshima, S., K. A. Frey, N. L. Foster and D. E. Kuhl (1995). "Preserved pontine glucose metabolism in Alzheimer disease: a reference region for functional brain image (PET) analysis." <u>J Comput Assist Tomogr</u> **19**(4): 541-547.
- Minoshima, S., R. A. Koeppe, K. A. Frey and D. E. Kuhl (1994). "Anatomic standardization: linear scaling and nonlinear warping of functional brain images." J Nucl Med **35**(9): 1528-1537.

- Morris, J. C. (1993). "The Clinical Dementia Rating (CDR): current version and scoring rules." Neurology **43**(11): 2412-2414.
- Morris, J. C., C. Ernesto, K. Schafer, M. Coats, S. Leon, M. Sano, L. J. Thal and P. Woodbury (1997). "Clinical dementia rating training and reliability in multicenter studies: the Alzheimer's Disease Cooperative Study experience." Neurology **48**(6): 1508-1510.
- Petersen, R. C., R. Doody, A. Kurz, R. C. Mohs, J. C. Morris, P. V. Rabins, K. Ritchie, M. Rossor, L. Thal and B. Winblad (2001). "Current concepts in mild cognitive impairment." <u>Arch Neurol</u> **58**(12): 1985-1992.
- Pontiroli, A. E., M. Alberetto, A. Secchi, G. Dossi, I. Bosi and G. Pozza (1982). "Insulin given intranasally induces hypoglycaemia in normal and diabetic subjects." <u>Br Med J (Clin Res Ed)</u> **284**(6312): 303-306.
- Reger, M. A., G. S. Watson, W. H. Frey, 2nd, L. D. Baker, B. Cholerton, M. L. Keeling, D. A. Belongia, M. A. Fishel, S. R. Plymate, G. D. Schellenberg, M. M. Cherrier and S. Craft (2006). "Effects of intranasal insulin on cognition in memory-impaired older adults: modulation by APOE genotype." Neurobiol Aging **27**(3): 451-458.
- Reger, M. A., G. S. Watson, P. S. Green, L. D. Baker, B. Cholerton, M. A. Fishel, S. R. Plymate, M. M. Cherrier, G. D. Schellenberg, W. H. Frey and S. Craft (2008). "Intranasal insulin administration dose-dependently modulates verbal memory and plasma amyloid-beta in memory-impaired older adults." <u>Journal of Alzheimers Disease</u> **13**(3): 323-331.
- Reger, M. A., G. S. Watson, P. S. Green, C. W. Wilkinson, L. D. Baker, B. Cholerton, M. A. Fishel, S. R. Plymate, J. C. Breitner, W. DeGroodt, P. Mehta and S. Craft (2008). "Intranasal insulin improves cognition and modulates beta-amyloid in early AD." <u>Neurology</u> **70**(6): 440-448.
- Rivera, E. J., A. Goldin, N. Fulmer, R. Tavares, J. R. Wands and S. M. de la Monte (2005). "Insulin and insulin-like growth factor expression and function deteriorate with progression of Alzheimer's disease: link to brain reductions in acetylcholine." J Alzheimers Dis 8(3): 247-268.
- Rubin, D. B. (1987). <u>Multiple Imputation for Nonresponse in Surveys</u>. Hoboken, New Jersey, John Wiley & Sons, Inc.
- Sakane, T., M. Akizuki, Y. Taki, S. Yamashita, H. Sezaki and T. Nadai (1995). "Direct drug transport from the rat nasal cavity to the cerebrospinal fluid: the relation to the molecular weight of drugs." <u>J</u> Pharm Pharmacol **47**(5): 379-381.
- Sano, M., R. Raman, J. Emond, R. G. Thomas, R. Petersen, L. S. Schneider and P. S. Aisen (2011). "Adding Delayed Recall to the Alzheimer Disease Assessment Scale is Useful in Studies of Mild Cognitive Impairment But Not Alzheimer Disease." <u>Alzheimer Dis Assoc Disord</u> **25**(2): 122-127. Scheen AJ. Sodium-glucose cotransporter type 2 inhibitors for the treatment of type 2 diabetes mellitus. Nat Rev Endocrinol. 2020 Oct;16(10):556-577. doi: 10.1038/s41574-020-0392-2. Epub 2020 Aug 27. PMID: 32855502.
- Selkoe, D. J. (2008). "Soluble oligomers of the amyloid beta-protein impair synaptic plasticity and behavior." <u>Behav Brain Res</u> **192**(1): 106-113.
- Shipley, M. T. (1985). "Transport of molecules from nose to brain: transneuronal anterograde and retrograde labeling in the rat olfactory system by wheat germ agglutinin-horseradish peroxidase applied to the nasal epithelium." <u>Brain Res Bull</u> **15**(2): 129-142.
- Stockhorst, U., D. de Fries, Y. Schottenfeld-Naor, A. Huebinger, H. J. Steingrueber and W. A. Scherbaum (Submitted for publication). "Intranasally administered insulin and its CNS effects in healthy humans: unconditioned and conditioned responses."
- Stockhorst, U., D. de Fries, H. J. Steingrueber and W. A. Scherbaum (2004). "Insulin and the CNS: effects on food intake, memory, and endocrine parameters and the role of intranasal insulin administration in humans." <a href="https://example.com/Physiol Behav">Physiol Behav</a> 83(1): 47-54.
- Talairach, J. and P. Tournoux (1988). <u>Co-planar stereotaxic atlas of the human brain: 3-dimensional proportional system: an aproach to cerebral imaging</u>. New York, New York, Thieme Medical Publishers.
- Thorne, R. G., C. R. Emory, T. A. Ala and W. H. Frey, 2nd (1995). "Quantitative analysis of the olfactory pathway for drug delivery to the brain." <u>Brain Res</u> **692**(1-2): 278-282.

Thorne, R. G., G. J. Pronk, V. Padmanabhan and W. H. Frey, 2nd (2004). "Delivery of insulin-like growth factor-I to the rat brain and spinal cord along olfactory and trigeminal pathways following intranasal administration." <u>Neuroscience</u> **127**(2): 481-496.

Townsend, M., T. Mehta and D. J. Selkoe (2007). "Soluble Abeta inhibits specific signal transduction cascades common to the insulin receptor pathway." J Biol Chem **282**(46): 33305-33312.

Weiss, P. and Y. Holland (1967). "Neuronal dynamics and axonal flow, ii. The olfactory nerve as model test object." Proc Natl Acad Sci U S A **57**(2): 258-264.

Worsley, K. J., A. C. Evans, S. Marrett and P. Neelin (1992). "A three-dimensional statistical analysis for CBF activation studies in human brain." J Cereb Blood Flow Metab **12**(6): 900-918.

Zhao, L., B. Teter, T. Morihara, G. P. Lim, S. S. Ambegaokar, O. J. Ubeda, S. A. Frautschy and G. M. Cole (2004). "Insulin-degrading enzyme as a downstream target of insulin receptor signaling cascade: implications for Alzheimer's disease intervention." <u>J Neurosci</u> **24**(49): 11120-11126.

Zhao, W. Q. and M. Townsend (2009). "Insulin resistance and amyloidogenesis as common molecular foundation for type 2 diabetes and Alzheimer's disease." Biochim Biophys Acta 1792(5): 482-496. Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS™ sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID: 22250775; PMCID: PMC3261577.

Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID: 11556941; PMCID: PMC1495268.

Spitzer RL, Kroenke K, Williams JB, Löwe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID: 16717171.